Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes (TECOS trial)

NCT03936062

December 27, 2019

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes (TECOS trial)

#### 1.2 <u>Intended aim(s)</u>

TECOS primarily tested the hypothesis that sitagliptin, when used as part of usual diabetes care, is non-inferior to usual care without sitagliptin with regard to the risk of significant confirmed cardiovascular outcomes.

### 1.3 Primary endpoint for replication and RCT finding

Composite of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, or hospitalization for unstable angina

### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Power of 90% for the test of noninferiority (hazard ratio, 1.00). For superiority, 1,300 patients with a primary composite cardiovascular outcome would provide a power of approximately 81% to determine the superiority of sitagliptin over placebo (hazard ratio, 0.85).

### 1.5 Primary trial estimate targeted for replication

HR = 0.98 (95% CI, 0.88 - 1.09) comparing sitagliptin to placebo (Green et al., 2015)

#### 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

### 3. Data Source(s)

United/Optum, MarketScan, Medicare

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

### **Design Diagram – TECOS TRIAL REPLICATION**



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, cohort study design comparing sitagliptin to the 2nd generation sulfonylurea (SU) antidiabetic class as a proxy for placebo. 2nd generation SUs are not known to have an impact on the outcome of interest. In addition, SUs were the most frequent background treatment in TECOS (after metformin), and both DPP4i and SUs are preferentially prescribed to similarly older patients in the real world (Patorno et al., 2019). The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of sitagliptin or a comparator drug (cohort entry date). Follow-up for the outcome (4P-MACE), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during the study.

### 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

#### 5.2.1 Eligible cohort entry dates

Market availability of sitagliptin in the U.S. started on October 17, 2006.

- For Marketscan: October 17, 2006-Dec 2017 (end of data availability).
- For Medicare: Jan 1, 2012-Dec 31, 2017 (start- end of data availability).
- For Optum: October 17, 2006-March 31, 2019 (end of data availability).

### 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

## 5.3 Flowchart of the study cohort assembly

| Optum | Marketscan | Medicare* |
|-------|------------|-----------|
|-------|------------|-----------|

| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
|---|---|---|---|---|---|---|
| All patients | | 74,864,884 | | 191,990,035 | | 23,466,175 |
| Patients who used exposure or a reference between <b>17 Oct 2006</b> to Dec 2017 (for Marketscan)/March 2019 (for Optum) and 01 January 2012-December 2017 for Medicare | -72908924 | 1,955,960 | -<br>188954110 | 3,035,925 | -19512001 | 3,954,174 |
| Excluded due to insufficient enrollment | -260546 | 1,695,414 | -374862 | 2,661,063 | -1094721 | 2,859,453 |
| Excluded due to prior use of referent | -1135398 | 560,016 | -1658570 | 1,002,493 | -1745525 | 1,113,928 |
| Excluded due to prior use of exposure | -237943 | 322,073 | -531814 | 470,679 | -511933 | 601,995 |
| Excluded because patient qualified in >1 exposure category | -1,240 | 320,833 | -3,027 | 467,652 | -1,510 | 600,485 |
| Excluded based on Age | -14 | 320,819 | 0 | 467,652 | 0 | 600,485 |
| Excluded based on Gender | -32 | 320,787 | 0 | 467,652 | 0 | 600,485 |
| Excluded based on Inclusion 1- DM Type 2 with ICD-10 | -31605 | 289,182 | -73914 | 393,738 | -11767 | 588,718 |
| Excluded based on Inclusion 1- Continuous use of Metformin, pioglitazone, or a sulfonylurea, or stable dose of insulin for past 3 months | -31597 | 257,585 | -50189 | 343,549 | -61901 | 526,817 |
| Excluded based on Inclusion 2- At least 2 outpatient visits in prior year | -533 | 257,052 | -1,385 | 342,164 | -412 | 526,405 |
| Excluded based on Inclusion 3- Age >=50 AND History of a major clinical manifestation of coronary artery disease/Ischemic cerebrovascular disease | -101729 | 155,323 | -167085 | 175,079 | -88675 | 437,730 |
| Excluded based on Exclusion 1- history of type 1 diabetes mellitus or a history of ketoacidosis | -3282 | 152,041 | -3487 | 171,592 | -9452 | 428,278 |
| Excluded based on Exclusion 2- ≥2 hospitalizations for severe Hypoglycemia in prior year | -21 | 152,020 | -39 | 171,553 | -318 | 427,960 |
| Excluded based on Exclusion 3- DPP-4 i, GLP-1, or a thiazolidinedione other than pioglitazone within past 3 months | -1711 | 150,309 | -1979 | 169,574 | -4416 | 423,544 |
| Excluded based on Exclusion 4- Cirrhosis of liver | -506 | 149,803 | -316 | 169,258 | -1,388 | 422,156 |
| Excluded based on Exclusion 7-Pregnancy | -8 | 149,795 | -7 | 169,251 | -13 | 422,143 |
| Excluded based on Exclusion 8- CCI 180days >=10 | -2092 | 147,703 | -1029 | 168,222 | -10402 | 411,741 |
| Final cohort | | 147,703 | | 168,222 | | 411,741 |

<sup>\*</sup> Medicare database includes only patients ≥65 years of age with at least one diagnosis for diabetes, heart failure, or stroke.

## 6. Variables

## 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is initiation of sitagliptin. Initiation will be defined by no use of sitagliptin or a comparator in the prior 6 months before treatment initiation (washout period).

#### Comparator agents:

- Initiators of sitagliptin will be compared to initiators of
  - o 2nd generation sulfonylureas

Because sitagliptin and comparators are frequently used as second or third line treatments of T2DM, we expect it to be unlikely that sitagliptin and comparators are initiated in patients with substantially different baseline risk for proposed outcomes.

#### 6.2 Preliminary covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B). These covariates are based on those used by Patorno et al. (2019).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Primary Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- <u>Primary outcome</u>: 4-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or CV mortality; as well as each individual component:
- Secondary outcomes: Individual MACE components:
  - o Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  - o Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  - Hospital admission for ACS/unstable angina
  - o All-cause mortality/CV mortality:
    - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in commercial databases
    - Information on CV mortality through data linkage with the National Death Index (NDI) will only become available at a later date for Medicare and will be used in secondary analyses.

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

1. Severe hypoglycemia (we expect to see protective effect; American Diabetes Association, 2018)

#### **Control outcome definitions**

| Outcome | Hospital Discharge Code(s) | Comments |
|---|---|---|
| Severe hypoglycemia | Severe hypoglycemia Any-position ED or primary inpatient ICD-9 diagnosis: 251.0, 251.1x, 251.2x, or 250.8x. Outcomes identified by 250.8x are not included if they co-occur with one of the following diagnoses: 259.8, 272.7, 681.xx, 682.xx, 686.9, 707.1x, 707.2x, 707.8, 707.9, 709.3, 730.0x, 730.1x, 730.2x, 731.8 | Note- The corresponding ICD-10 codes will be used also |

## 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of liraglutide and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (sitagliptin and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from an exposure to a comparator or any other agent in the comparator class and vice versa (e.g. switching from glimepiride to glipizide would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - An added treatment that is not part of the exposure or comparator group does not fulfill this criterion (e.g. if a sitagliptin user adds insulin, he or she does not get censored at the time of insulin augmentation)

For the ITT analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

### 7. Initial Feasibility Analysis

### Aetion report links:

Optum: https://bwh-dope.aetion.com/#/projects/details/640/results/26047/result/0
Marketscan: https://bwh-dope.aetion.com/#/projects/details/638/results/26040/result/0
Medicare: https://bwh-dope.aetion.com/#/projects/details/639/results/26043/result/0

Date conducted: Sep 30, 2018

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### Aetion report links:

Optum: https://bwh-dope.aetion.com/#/projects/details/640/results/26049/result/0
Marketscan: https://bwh-dope.aetion.com/#/projects/details/638/results/26050/result/0
Medicare: https://bwh-dope.aetion.com/#/projects/details/639/results/26051/result/0

Date conducted: Sep 30, 2018

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated in the subsequent sections, after incorporating feedback and refining the protocol.

| Reviewed by PI: | Jessica M. Franklin | Date reviewed: | 10/26/18 |
|-------------------------|---------------------|----------------|----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 12/11/18 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

### 9. Balance Assessment after PS matching

## Aetion report links (Sitagliptin vs. 2<sup>nd</sup> generation SUs):

Optum: https://bwh-dope.aetion.com/projects/details/640/results/44780/result/0
Marketscan: https://bwh-dope.aetion.com/projects/details/638/results/44781/result/0
Medicare: https://bwh-dope.aetion.com/projects/details/639/results/45413/result/0

Date conducted: 11/18/2019 (Medicare 11/30/2019)

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 7,596 (2.17%) | 4,072 (2.33%) | 3,524 (2.02%) |
| Start of an additional exposure | 22,929 (6.56%) | 6,881 (3.94%) | 16,048 (9.18%) |
| End of index exposure | 210,496 (60.23%) | 104,902 (60.03%) | 105,594 (60.43%) |
| Specified date reached | 36,338 (10.40%) | 19,668 (11.26%) | 16,670 (9.54%) |
| End of patient enrollment | 33,356 (9.54%) | 17,150 (9.81%) | 16,206 (9.27%) |
| Switch to other SUs (for censoring) + nursing home admission | 38,761 (11.09%) | 22,065 (12.63%) | 16,696 (9.55%) |

• Report follow-up time by treatment group.

| | N | Median Follow-Up Time (Days) [IQR] | |
|---|---|---|---|
| Patient Group | Optum | Marketscan | Medicare |
| Overall Patient Population | 118 [58-270] | 120 [58-300] | 118 [58-297] |
| Referent | 118 [58-295] | 121 [58-316] | 121 [58-316] |
| Exposure | 118 [58-246] | 118 [58-279] | 118 [58-279] |

• Report overall risk of the primary outcome.

| | Optum | Marketscan | Medicare |
|-------------------------|-------|------------|----------|
| Risk per 1,000 patients | 29.17 | 37.73 | 62.67 |

#### 10. Final Power Assessment

#### Date conducted:

- Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).
  - o Pooled

| Non-inferiority Analysis | | Superiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 174,738 | Reference | 174,738 |
| Exposed | 174,738 | Exposed | 174,738 |
| Risk per 1,000 patients | 43.19 | Risk per 1,000 patients | 43.19 |
| Assumed HR from RCT | 1 | Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 1.3 | | |
| Number of events expected | 15093.86844 | Number of events expected | 15093.86844 |
| Power | 1 | Power | 1 |

## o Optum

| Non-inferiority Analysis | | Superiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 29,727 | Reference | 29,727 |
| Exposed | 29,727 | Exposed | 29,727 |
| Risk per 1,000 patients | 29.17 | Risk per 1,000 patients | 29.17 |
| Assumed HR from RCT | 1 | Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 1.3 | | |
| Number of events expected | 1734.27318 | Number of events expected | 1734.27318 |
| Power | 0.999770031 | Power | 0.92278468 |

## Marketscan

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

| Non-inferiority Analysis | | Superiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 42,600 | Reference | 42,600 |
| Exposed | 42,600 | Exposed | 42,600 |
| Risk per 1,000 patients | 37.73 | Risk per 1,000 patients | 37.73 |
| Assumed HR from RCT | 1 | Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 1.3 | | |
| Number of events expected | 3214.596 | Number of events expected | 3214.596 |
| Power | 0.99999978 | Power | 0.995942377 |

## Medicare

| Non-inferiority Analysis | | Superiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 102,411 | Reference | 102,411 |
| Exposed | 102,411 | Exposed | 102,411 |
| Risk per 1,000 patients | 62.67 | Risk per 1,000 patients | 62.67 |
| Assumed HR from RCT | 1 | Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| Non-inferiority margin | 1.3 | | |
| Number of events expected | 12836.19474 | Number of events expected | 12836.19474 |
| Power | 1 | Power | 1 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of

advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/9/19 |
|-------------------------|------------------|----------------|----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 12/20/19 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns: 12/20/19

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.

### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

Aetion report name:

<u>Date conducted:</u>

### 13.1 For primary analysis:

• In the PS-matched cohort from Section 9, calculate the HR for each outcome for sitagliptin versus 2<sup>nd</sup> generation SU patients using a Cox proportional hazards model.

#### 13.2 For secondary analyses:

• In both pre-matched cohorts, perform asymmetrical trimming to remove patients with PS values below the 2.5<sup>th</sup> percentile of treated patients and above the 97.5<sup>th</sup> percentile of untreated patients. In the trimmed cohort, calculate the HR for canagliflozin versus referent patients using a Cox proportional hazards model, adjusting for deciles of the PS.

#### 14. Requested Results

### 14.1 Results from primary and secondary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Primary analysis | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

#### 15. References

American Diabetes Association. 8. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018;41(Suppl 1):S73-S85. doi:10.2337/dc18-S008.

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. **page** 177

Green JB, Bethel MA, Armstrong PW, Buse JB, Engel SS, Garg J, Josse R, Kaufman KD, Koglin J, Korn S, Lachin JM. Effect of sitagliptin on cardiovascular outcomes in type 2 diabetes. New England Journal of Medicine. 2015; 373(3):232-42.

Effectiveness research with Real World Data to support FDA's regulatory decision making

Patorno E, Pawar A, Franklin JM, et al. Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. Circulation. 2019; in press. (https://www.ahajournals.org/doi/pdf/10.1161/CIRCULATIONAHA.118.039177)

| # | TECOS trial definitions | Implementation in routine care | Please see the following Google Drive for further deta<br>https://drive.google.com/open?id=1WD618wryw | |
|---|---|---|---|---|
| | Trial details- 2b- Failed S with NI- P | io label change | ICD-10 codes are not listed in this document because of excel cell size limitati code lists will be available in the above Google Drive Folder (link above). ICD-9 macro that implements forward/backward mapping based of https://www.nber.org/data/icd9-icd-10-cm-and-pcs-crosswa | to ICD-10 code conversions were completed using a SAS on the CMS ICD-9 to ICD-10 mapping: |
| | EXPOSURE vs. COMPAR | ISON | Reference/Rationale | Color coding |
| | Sitagliptin versus placebo | Sitagliptin vs. 2nd generation sulfonylureas | | Criteria |
| | PRIMARY OUTCOM | | | Adequate mapping in claims |
| | The primary cardiovascular outcome was a composite of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, or hospitalization for unstable angina. HR 0.98; 95% CI, 0.88 to 1.09; P<0.001 | Measured 1 days after drug initiation in diagnosis position specified below and inpatient care setting: Inpatient mortality/MI/Stroke/Angina — For ACS/unstable angina Any diagnosis position in inpatient care setting Discharge diagnosis ICD-9 411.xx For MI Any diagnosis position in inpatient care setting ICD-9 Dx 410.X (acute myocardial infarction) excluding 410.x2 (subsequent episode of care) For stroke Primary diagnosis position in inpatient care setting ICD-9 discharge diagnosis: 430.xx Subarachnoid hemorrhage (SAH) 431.xx Intracerebral hemorrhage (ICH) 433.x1 Occlusion and stenosis of precerebral arteries with cerebral infarction 434.xx (excluding 434.xX) Occlusion and stenosis of cerebral arteries with cerebral infarction 436.x Acute, but ill-defined cerebrovascular events Mortality-See Mortality Sheet. | For MI: →PPV 94% in Medicare claims data [Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. American heart journal 2004;148:99-104.] →PPV 88.4% in commercially-insured population [Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. Pharmacoepidemiology and Drug Safety 2010;19:596-603.] For stroke: PPV 188.5% or higher for ischemic stroke PPV ranging from 80% to 98% for hemorrhagic stroke →[Andrade SE, Harrold LR, Tjia J, et al. A systematic review of validated methods for identifying ereerbovascular accident or transient ischemic attack using administrative data. Pharmacoepidemiology and Drug Safety 2012;21 Suppl 1:100-28.] →[Tirschwell DL, Longstreth WT, Jr. Validating administrative data in stroke research. Stroke; a journal of cerebral circulation 2002;33:2465-70.] →[Roumie CL, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsaguel, Griffin MR. Validation of ICO-9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. Pharmacoepidemiology and drug safety 2008;17:20-6.] | Intermediate mapping in claims |
| | INCLUSION CRITERIA | | | Poor mapping or cannot be measured in claims |
| | Patient has T2DM with HbA1c of≥6.5% (48 mmol/mol) and ≤8.0% (64 mmol/mol). HbA1c must be documented within 3 months prior to study enrollment, while receiving either: | Measured 180 days prior to drug initiation any diagnosis position in inpatient or outpatient care settings: Patients with a diagnosis of T2DM (ICD-9 Dx code of 250.x0 or 250.x2; ICD-10 Dx code of E11.x) in the 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi:10.1161/CIRCULATIONAHA.118.039177 | Can't be measured in claims but not important for the analysis |
| 1 | <ul> <li>Metformin, pioglitazone, or a sulfonylurea as monotherapy or any dual combination of metformin, pioglitazone,<br/>or a sulfonylurea continuously without alteration in dose for at least 3 months. Note: patients who have received<br/>insulin for only a short period (i.e. less than 14 days) during a hospitalization or for the management of acute illness<br/>will not be excluded for that reason.</li> </ul> | Measured 91 days prior to drug initiation as any dispensing of one of the following drugs:<br>Metformin, pioglitazone, or a sulfonylurea (monotherapy or any dual combination) | | |
| | • A stable dose of insulin (±20% of the scheduled total daily insulin dose) either alone or in combination with a stable dose of metformin for at least 3 months. The use of supplemental/sliding scale insulin during the prior 3 months is permissible, as long as the total daily insulin dose is within ±20% of the scheduled total daily insulin dose. Note: Patients who have required modification of their usual daily insulin dose for a short period (b14 days) during a hospitalization or for the management of acute illness will not be excluded for that reason. | Measured 91 days prior to drug initiation as any dispensing of insulin (Please see AHA therapies sheet for full definition). | | |
| | Patient is able to see a usual care provider at least twice per year. | Measured 365 days prior to drug initiation as any 2 claims in outpatient care setting | | |
| 2 | Patient is ≥50 years of age with pre-existing vascular disease, defined as having any one of the following: | Patient is ≥50 years of age measured on day of drug initiation | I | Ī |

| 3a | History of a major clinical manifestation of coronary artery disease (i.e., Ml, surgical or percutaneous [balloon and/or stent] coronary revascularization procedure, or coronary angiography showing at least one stenosis 250% in a major epicardial artery or branch vessel); | Measured 365 days prior to drug initiation in any diagnosis/procedure position and care setting defined below: Inpatient or outpatient Acute MI: 410.xx, Inpatient or outpatient Old MI: 412.xx Also include 414.xx (Inpatient or outpatient) PTCA: Inpatient CPT-4: 92973, 92982, 92984, 92995, 92996, 92920 – 92921, 92924 – 92925, 92937, 92938, 92941, 92943, 92944 OR — Inpatient or outpatient ICD-9 procedure: 00.66, 36.01, 36.02, 36.03, 36.05, 36.09 Stenting: Inpatient CPT-4: 92980, 92981, 92928 – 92929, 92933 – 92934 OR — Inpatient or outpatient ICD-9 procedure: 36.06, 36.07 CABG: Inpatient CPT-4: 33510 – 33536, 33545, 33572. OR — Inpatient or outpatient ICD-9 procedure: 36.1x, 36.2x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
|---|---|---|---|
| 3b | Ischemic cerebrovascular disease, including: | | |
| | • History of ischemic stroke. Strokes not known to be hemorrhagic will be allowed as part of this criterion; | Measured 365 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting: Ischemic stroke (w and w/o mention of cerebral infarction)- 433.xx, 434.xx, 436.xx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | - History of carotid arterial disease as documented by ≥50% stenosis documented by carotid ultrasound, magnetic resonance imaging (MRI), or angiography, with or without symptoms of neurologic deficit. | Measured 365 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting: Occlusion and stenosis of carotid artery without mention of cerebral infarction 433.10 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | Atherosclerotic peripheral arterial disease, as documented by objective evidence such as amputation due to vascular disease, current symptoms of intermittent claudication confirmed by an ankle brachial pressure index or toe brachial pressure index less than 0.9, or history of surgical or percutaneous revascularization procedure. | Measured 365 days prior to drug initiation in any diagnosis/procedure position and inpatient or outpatient care setting: Peripheral arterial stenting or surgical revascularization ICD-9 39,25, 39,50, 39,99. Lower extremity amputation ICD-9 diagnosis: V49,7x ICD-9 procedure: 84,10-84,18 CPT: 27590, 27591, 27592, 27880, 27881, 27882, 27884, 27886, 27888, 27889, 28800, 28805, 28810, 28820, 28825 Ankle brachial pressure index <0.9 ICD-9 440.21 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/pmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | Female patients agree to use an effective method of contraception or must not otherwise be at risk of becoming pregnant. | Since this is an inclusion criteria, it's difficult to implement the contraceptive use requirement here, but we have pregnancy as an exclusion criteria later, so this requirement is implemented then. | |
| | Patient understands the study procedures, alternative treatments available, and the risks involved with the study, and voluntarily agrees to participate by providing written informed consent. | N/A | |
| | Patient agrees to provide permission to obtain all medical records necessary for complete data ascertainment during the follow-up period. | N/A | |
| | EXCLUSION CRITERI | A | |
| | 1. Patient has a history of type 1 diabetes mellitus or a history of ketoacidosis. | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting: DM type 1-At least 1 inpatient or outpatient ICD-9 Dx code of 250.x1 or 250.x3 or ICD-10 Dx code of £10.x in the 6 months prior to drug initiation. Ketoacidosis 250.1x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |

| 2 hy | atient has a history of ≥ <b>2 episodes of severe hypoglycemia during the 12 months</b> prior to enrollment. Severe<br>ypoglycemia (hypoglycemia requiring assistance) refers to instances in which the patient was sufficiently<br>soriented or incapacitated as to require help from another individual or from medical personnel (whether or not<br>is assistance was actually provided). | Measured 365 days prior to drug initiation in any diagnosis position and inpatient care setting: 251.1x, 251.20, 962.30 Also, 250.8x as long as none of the following codes are co-occurring diagnoses (i.e. same day): 259.8, 272.7,681.xx, 682.xx, 686.9x, 707.xx, 709.3, 730.0-730.2, 731.8 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
|---|---|---|---|
| 3 vi | atient has taken an approved or investigational DPP-4 inhibitor agent (eg. sitagliptin, alogliptin, saxagliptin, or<br>Idagliptin), GLP-1 analogues (eg. exenatide, exenatide LAR, or liraglutide), or a thiazolidinedione other than<br>oglitazone within the past 3 months. | Measured 91 days prior to drug initiation as a dispensing of one of the following drugs: DDP-4,<br>GLP-1, or a thiazolidinedione (other than pioglitazone). Please see full definition in the AHA<br>therapies sheet. | |
| <b>4</b> Pa | atient has cirrhosis of the liver, as assessed by medical history. | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or<br>outpatient care setting:<br>Liver cirrhosis-571.2, 571.5, 571.6 | Karagozian R et al. "Obesity paradox in advanced liver disease: obesity is associated with lower mortality in hospitalized patients with cirrhosis." Liver int. 2016 Oct; 1450-6. doi: 10.1111/liv.13137. Epub 2016 May 4. |
| | atient is enrolled in another experimental protocol which involves the use of an investigational drug or device, or a intervention that would interfere with the conduct of the trial. | N/A | |
| 6 Pa | atient has a <b>planned or anticipated</b> revascularization procedure. | N/A | |
| <b>7</b> Pr | regnancy or planned pregnancy during the trial period. | | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | atient has medical history that indicates a life expectancy of <2 years or might limit the individual's ability to take ial treatments for the duration of the study. | Measured 180 days prior to drug initiation: Exclude patients with a combined comorbidity score >=10 | Gagne, Josh J et. al. "A combined comorbidity score predicted mortality in elderly patients better than existing scores." J Clin Epidemiol. 2011 Jul;64(7):749-59. doi: 10.1016/j.jclinepi.2010.10.004. Sun, Jenny W et. al. "Validation of the Combined Comorbidity Index of Charlson and Elixhauser to Predict 30-Day Mortality Across ICD-9 and ICD-10." Med Care. 2018 Sep;56(9):812. doi: 10.1097/MLR.000000000000954. |
| 9 in | atient has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance which,<br>the opinion of the investigator or coordinator, might pose a risk to the patient, make participation not in the<br>stient's best interest, confound the results of the study (eg. if patient cannot comply with requirements of the<br>udy), or interfere with the patient's participation for the full duration of the study. | N/A | |
| 10 | atient has an estimated GFR (calculated based on serum creatinine via the MDRD formula) of b30 mL/ min per 73 m2. | N/A | |
| | atient has a known allergy or intolerance to sitagliptin. | N/A | |
| 12 Pa | atient has previously been enrolled in the trial. | N/A | |

| Trial ID | |
|---|---|
| Trial Name (with web links) | TECOS |
| Trial Name (with pdf links) | |
| <u>NCT</u> | NCT00790205 |
| Trial category | |
| Therapeutic Area | Endocrinology |
| RCT Category | 2b- Failed S with NI- No label change |
| <b>Brand Name</b> | |
| <b>Generic Name</b> | Sitagliptin |
| Sponsor | Merck Sharp & Dohme Corp. |
| <u>Year</u> | 2015 |
| | Composite of cardiovascular death, nonfatal myocardial |
| | infarction, nonfatal stroke, or hospitalization for unstable |
| Measurable endpoint | angina |
| <u>Exposure</u> | Sitagliptin |
| <u>Comparator</u> | Placebo |
| <u>Population</u> | |
| <u>Trial finding</u> | HR 0.98; 95% CI, 0.88 to 1.09; P<0.001 |
| <u>Notes</u> | |
| No. of Patients | |
| Non-inferiority margin | HR = 1.30 |
| Assay Sens. Endpoint | |
| Assay Sens. Finding | |
| <u>Ajinkya comments</u> | |
| | power of approximately 81% to determine the |
| Power | superiority of sitagliptin over placebo (hazard ratio, 0.85) |
| Blinding | |
| Statistical Method | |
| Approval indication | |

### Mortality-Dependent on data source.

1. All-cause mortality / inpatient mortality Identified using the vital status file-

#### Medicare

Identified using the discharge status codes-

#### Optum-

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

#### Truven-

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)
- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)

- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

## 2. CV mortality

Information on CV mortality through data linkage with the National Death Index (NDI) will be available for Medicare and Optum Clinformatics at a later date. We will conduct secondary analyses using CV mortality at that time.

| Antidiabetic class | Specific agent | Notes |
|---|---|---|
| | Canagliflozin | Approved 3/29/2013 |
| SCI T2 :1:1:1: | Dapagliflozin | |
| SGL 12-innibitors | Empagliflozin | |
| | Ertugliflozin | Approved Dec 21, 2017 |
| | Glimepiride | |
| 2 <sup>nd</sup> generation sulfonylureas | Glipizide | |
| | Glyburide | |
| | Alogliptin | |
| IDDD 4 in Lil. it and | Linagliptin | |
| DPP-4 innibitors | Saxagliptin | |
| | Sitagliptin | |
| | Exenatide | |
| | Liraglutide | |
| GLT2-inhibitors In generation sulfonylureas PP-4 inhibitors LP-1 receptor agonist (GLP1-RA) | Albiglutide | Approved April 15, 2014 and discontinued July 26, 2017 |
| , | Dulaglutide | Approved Sep 18, 2014 |
| | Lixisenatide | Approved July 28, 2016 |
| | Semaglutide | Approved Dec 5, 2017 |
| | Insulin Aspart | |
| | Insulin Aspart/Insulin Aspart Protamine | |
| | Insulin Degludec | |
| | Insulin Detemir | |
| | Insulin Glargine | |
| | Insulin Glulisine | |
| Insulin | Insulin human isophane (NPH) | |
| | Insulin human regular (search with NPH, don't want bf-pk) | |
| | Insulin human regular/ Insulin human isophane (NPH) | |
| | Insulin Lispro | |
| | Insulin Lispro/Insulin Lispro Protamine | |
| | Pioglitazone | † |

| Uiitazuiies | Rosiglitazone |
|------------------------------------------|----------------|
| leglitinides lpha-glucosidase inhibitors | Nateglinide |
| Megnunides | Repaglinide |
| lpha-glucosidase inhibitors | Acarbose |
| Alpha-glucosidase illinoitors | Miglitol |
| Pramlintide | Pramlintide |
| | Acetohexamide |
| pha-glucosidase inhibitors | Chlorpropamide |
| generation suffonytureas | Tolazamide |
| | Tolbutamide |

## Pregnancy Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION

- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION

- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS



Table 1: Sitagliptin vs 2nd Generation Sulfonylureas

| Unmatched | Unmatched | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| F | Optun | n I | MarketS | can | Medicare | | | POOLED | |
| - | Reference- 2nd | | Reference-2nd | | Reference-2nd | Exposure- | Reference-2nd | | |
| Variable | Generation SUs | Exposure-Sitagliptin | Generation SUs | Exposure-Sitagliptin | Generation SUs | Sitagliptin | Generation SUs | Exposure-Sitagliptin | St. Diff. |
| Number of patients | 117,685 | 29,759 | 124,594 | 43,306 | 306,304 | 103,677 | 548,583 | 176,742 | |
| Age | | | | | | | | | |
| mean (sd) | 69.87 (9.37) | 69.12 (9.34) | 67.93 (10.74) | 66.24 (10.14) | 75.78 (7.53) | 75.65 (7.46) | 72.73 (8.76) | 72.24 (8.52) | 0.06 |
| median [IQR] | 70.00 [63.00, 77.00] | 69.00 [62.00, 76.00] | 66.00 [59.00, 77.00] | 64.00 [59.00, 74.00] | 75.00 [70.00, 81.00] 5 | .00 [70.00, 81.00] | 71.88 (8.76) | 71.29 (8.52) | 0.07 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 7,614 (6.5%) | 2,061 (6.9%) | 12,188 (9.8%) | 4,808 (11.1%) | 0 (0.0%) | 0 (0.0%) | 19,802 (3.6%) | 6,869 (3.9%) | -0.02 |
| 55 - 64; n (%) | 26,192 (22.3%) | 7,381 (24.8%) | 45,377 (36.4%) | 18,182 (42.0%) | 5,258 (1.7%) | 1,675 (1.6%) | 76,827 (14.0%) | 27,238 (15.4%) | -0.04 |
| 65 - 74; n (%) | 43,590 (37.0%) | 11,349 (38.1%) | 29,690 (23.8%) | 10,347 (23.9%) | 143,586 (46.9%) | 49,319 (47.6%) | 216,866 (39.5%) | 71,015 (40.2%) | -0.01 |
| >= 75; n (%) | 40,289 (34.2%) | 8,968 (30.1%) | 37,339 (30.0%) | 9,969 (23.0%) | 157,460 (51.4%) | 52,683 (50.8%) | 235,088 (42.9%) | 71,620 (40.5%) | 0.05 |
| Gender- | 70,996 (60.3%) | 16,783 (56.4%) | 78,953 (63.4%) | 26,549 (61.3%) | 159.873 (52.2%) | 49,637 (47.9%) | 309,822 (56.5%) | 92,969 (52.6%) | 0.08 |
| Males; n (%) | 70,996 (60.3%)<br>46,689 (39.7%) | 16,783 (56.4%) | 78,953 (63.4%)<br>45,641 (36.6%) | 26,549 (61.3%)<br>16,757 (38.7%) | 159,873 (52.2%)<br>146,431 (47.8%) | 49,637 (47.9%)<br>54,040 (52.1%) | 238,761 (43.5%) | 92,969 (52.6%)<br>83,773 (47.4%) | -0.08 |
| Females; n (%) Race without zero category | 40,089 (39.7%) | 12,3/0 (43.0%) | 43,041 (30.0%) | 10,/5/ (38./%) | 140,431 (47.8%) | 54,040 (52.1%) | 230,/01 (43.5%) | 03,//3 (4/.4%) | -0.08 |
| White; n (%) | N/A | N/A | N/A | N/A | 243,220 (79.4%) | 78,796 (76.0%) | 243,220 (79.4%) | 78,796 (76.0%) | 0.08 |
| wnite; n (%)<br>Black; n (%) | N/A | N/A<br>N/A | N/A<br>N/A | N/A | 35,871 (11.7%) | 12,037 (11.6%) | 35,871 (11.7%) | 12,037 (11.6%) | 0.08 |
| Asian; n (%) | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | N/A | 7,863 (2.6%) | 4,365 (4.2%) | 7,863 (2.6%) | 4,365 (4.2%) | -0.09 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 10,197 (3.3%) | 4,546 (4.4%) | 10,197 (3.3%) | 4,546 (4.4%) | -0.06 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 1,936 (0.6%) | 527 (0.5%) | 1,936 (0.6%) | 527 (0.5%) | 0.01 |
| Other/Unknown; n (%) | N/A | N/A | N/A | N/A | 7,217 (2.4%) | 3,406 (3.3%) | 7,217 (2.4%) | 3,406 (3.3%) | -0.05 |
| | | | .4 | .4 | , , ,, | -, (,-) | , | -, (- ,,-) | |
| Region- (lumping missing&other category with West) | | | | | | | | | |
| Northeast; n (%) | 11,989 (10.2%) | 4,227 (14.2%) | 19,997 (16.0%) | 9,324 (21.5%) | 53,453 (17.5%) | 24,496 (23.6%) | 85,439 (15.6%) | 38,047 (21.5%) | -0.15 |
| South; n (%) | 57,501 (48.9%) | 15,058 (50.6%) | 40,843 (32.8%) | 11,503 (26.6%) | 136,902 (44.7%) | 42,919 (41.4%) | 235,246 (42.9%) | 69,480 (39.3%) | 0.07 |
| Midwest; n (%) | 24,332 (20.7%) | 5,057 (17.0%) | 48,364 (38.8%) | 17,570 (40.6%) | 72,970 (23.8%) | 19,059 (18.4%) | 145,666 (26.6%) | 41,686 (23.6%) | 0.07 |
| West; n (%) | 23,863 (20.3%) | 5,417 (18.2%) | 14,184 (11.4%) | 4,488 (10.4%) | 42,979 (14.0%) | 17,203 (16.6%) | 81,026 (14.8%) | 27,108 (15.3%) | -0.01 |
| Unknown+missing; n (%) | N/A | N/A | 1,206 (1.0%) | 421 (1.0%) | N/A | N/A | 1,206 (1.0%) | 421 (1.0%) | 0.00 |
| CV Covariates | 78,804 (67.0%) | 19,763 (66.4%) | 79,177 (63.5%) | 27,756 (64.1%) | 208,853 (68.2%) | 70,050 (67.6%) | 366,834 (66.9%) | 117,569 (66.5%) | 0.01 |
| Ischemic heart disease; n (%) Acute MI; n (%) | 78,804 (67.0%) | 1,556 (5.2%) | 7,950 (6.4%) | 2,449 (5.7%) | 14,690 (4.8%) | 4,757 (4.6%) | 29,756 (5.4%) | 8,762 (5.0%) | 0.01 |
| ACS/unstable angina; n (%) | 6,453 (5.5%) | 1,610 (5.4%) | 7,950 (6.4%) | 2,520 (5.8%) | 12,974 (4.2%) | 4,714 (4.5%) | 26,516 (4.8%) | 8,762 (5.0%)<br>8,844 (5.0%) | -0.01 |
| Old MI; n (%) | 11,986 (10.2%) | 2,817 (9.5%) | 6,665 (5.3%) | 2,069 (4.8%) | 31,200 (10.2%) | 9,830 (9.5%) | 49,851 (9.1%) | 14,716 (8.3%) | 0.03 |
| Stable angina; n (%) | 9,950 (8.5%) | 2,606 (8.8%) | 8,129 (6.5%) | 3,044 (7.0%) | 22,435 (7.3%) | 8,273 (8.0%) | 40,514 (7.4%) | 13,923 (7.9%) | -0.02 |
| Coronary atherosclerosis and other forms of chronic | 3,550 (0.570) | 2,000 (0.070) | 5,125 (5.570) | 5,5 (7.070) | 22,133 (7.370) | 3,2,3 (3.370) | .0,52. (7.470) | 15,525 (7.570) | 0.02 |
| ischemic heart disease; n (%) | 74,752 (63.5%) | 18,866 (63.4%) | 75,286 (60.4%) | 26,621 (61.5%) | 201,279 (65.7%) | 67,394 (65.0%) | 351,317 (64.0%) | 112,881 (63.9%) | 0.00 |
| Other atherosclerosis with ICD10; n (%) | 3,467 (2.9%) | 858 (2.9%) | 3,167 (2.5%) | 1,108 (2.6%) | 10,599 (3.5%) | 3,723 (3.6%) | 17,233 (3.1%) | 5,689 (3.2%) | -0.01 |
| Previous cardiac procedure (CABG or PTCA or Stent) v4; n | | . , | | , , | | | | | |
| (%) | 4,865 (4.1%) | 1,125 (3.8%) | 6,743 (5.4%) | 2,291 (5.3%) | 7,210 (2.4%) | 2,586 (2.5%) | 18,818 (3.4%) | 6,002 (3.4%) | 0.00 |
| History of CABG or PTCA; n (%) | 18,909 (16.1%) | 4,629 (15.6%) | 9,546 (7.7%) | 3,482 (8.0%) | 60,080 (19.6%) | 19,148 (18.5%) | 88,535 (16.1%) | 27,259 (15.4%) | 0.02 |
| Any stroke; n (%) | 25,490 (21.7%) | 6,467 (21.7%) | 26,317 (21.1%) | 8,740 (20.2%) | 73,052 (23.8%) | 25,655 (24.7%) | 124,859 (22.8%) | 40,862 (23.1%) | -0.01 |
| Ischemic stroke (w and w/o mention of cerebral | | | | | | | | | |
| infarction); n (%) | 25,318 (21.5%) | 6,437 (21.6%) | 26,168 (21.0%) | 8,684 (20.1%) | 72,515 (23.7%) | 25,469 (24.6%) | 124,001 (22.6%) | 40,590 (23.0%) | -0.01 |
| Hemorrhagic stroke; n (%) | 785 (0.7%) | 181 (0.6%) | 821 (0.7%) | 273 (0.6%) | 2,062 (0.7%) | 741 (0.7%) | 3,668 (0.7%) | 1195 (0.7%) | 0.00 |
| TIA; n (%) | 5,153 (4.4%) | 1,294 (4.3%) | 5,539 (4.4%) | 1,696 (3.9%) | 14,598 (4.8%) | 5,155 (5.0%) | 25,290 (4.6%) | 8,145 (4.6%) | 0.00 |
| Other cerebrovascular disease; n (%) | 5,877 (5.0%) | 1,522 (5.1%) | 4,899 (3.9%) | 1,570 (3.6%) | 18,592 (6.1%) | 6,646 (6.4%) | 29,368 (5.4%) | 9,738 (5.5%) | 0.00 |
| Late effects of cerebrovascular disease; n (%) | 6,322 (5.4%) | 1,505 (5.1%) | 4,660 (3.7%) | 1,422 (3.3%) | 19,216 (6.3%) | 6,725 (6.5%) | 30,198 (5.5%) | 9,652 (5.5%) | 0.00 |
| Cerebrovascular procedure; n (%) | 548 (0.5%) | 95 (0.3%) | 658 (0.5%) | 185 (0.4%) | 1,139 (0.4%) | 370 (0.4%) | 2,345 (0.4%) | 650 (0.4%) | 0.00 |
| Heart failure (CHF); n (%) | 24,633 (20.9%) | 5,822 (19.6%) | 20,633 (16.6%) | 6,241 (14.4%) | 74,334 (24.3%) | 24,555 (23.7%) | 119,600 (21.8%) | 36,618 (20.7%) | 0.03 |
| Peripheral Vascular Disease (PVD) or PVD Surgery ; n (%) | 17,611 (15.0%) | 4,589 (15.4%) | 14,270 (11.5%) | 4,895 (11.3%) | 60,993 (19.9%) | 22,399 (21.6%) | 92,874 (16.9%) | 31,883 (18.0%) | -0.03 |
| Atrial fibrillation; n (%) | 17,961 (15.3%) | 4,302 (14.5%) | 16,153 (13.0%) | 5,109 (11.8%) | 64,943 (21.2%) | 21,134 (20.4%) | 99,057 (18.1%) | 30,545 (17.3%) | 0.03 |
| Other cardiac dysrhythmia; n (%) | 20,210 (17.2%) | 5,107 (17.2%) | 17,075 (13.7%) | 5,812 (13.4%) | 67,788 (22.1%) | 23,313 (22.5%) | 105,073 (19.2%) | 34,232 (19.4%) | -0.01 |
| Cardiac conduction disorders; n (%) | 6,876 (5.8%) | 1,676 (5.6%) | 5,401 (4.3%) | 1,770 (4.1%) | 24,291 (7.9%) | 7,964 (7.7%) | 36,568 (6.7%) | 11,410 (6.5%) | 0.01 |
| Other CVD; n (%) | 28,933 (24.6%) | 7,152 (24.0%) | 26,394 (21.2%) | 9,187 (21.2%) | 86,701 (28.3%) | 29,729 (28.7%) | 142,028 (25.9%) | 46,068 (26.1%) | 0.00 |
| Diabetes-related complications | / (//) | . , (/) | / (2/9) | -, (2/0) | ,(-3.370) | - / ( /0) | - :-, (:3/0) | , | 2.50 |
| Diabetic retinopathy; n (%) | 6,792 (5.8%) | 1,907 (6.4%) | 4,974 (4.0%) | 1,711 (4.0%) | 19,459 (6.4%) | 7,094 (6.8%) | 31,225 (5.7%) | 10,712 (6.1%) | -0.02 |
| | | | | | | | . , . , | | |
| Diabetes with other ophthalmic manifestations; n (%) | 543 (0.5%) | 145 (0.5%) | 3,717 (3.0%) | 1,300 (3.0%) | 7,490 (2.4%) | 2,860 (2.8%) | 11,750 (2.1%) | 4,305 (2.4%) | -0.02 |

| Retinal detachment, vitreous hemorrhage, vitrectomy; n | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (%) | 502 (0.4%) | 149 (0.5%) | 425 (0.3%) | 169 (0.4%) | 1,324 (0.4%) | 477 (0.5%) | 2,251 (0.4%) | 795 (0.4%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 687 (0.6%) | 173 (0.6%) | 814 (0.7%) | 289 (0.7%) | 1,636 (0.5%) | 625 (0.6%) | 3,137 (0.6%) | 1,087 (0.6%) | 0.00 |
| Occurrence of Diabetic Neuropathy ; n (%) | 21,372 (18.2%) | 5,846 (19.6%) | 13,374 (10.7%) | 4,906 (11.3%) | 61,487 (20.1%) | 22,354 (21.6%) | 96,233 (17.5%) | 33,106 (18.7%) | -0.03 |
| Occurrence of diabetic nephropathy with ICD10; n (%) | 17,094 (14.5%) | 4,492 (15.1%) | 6,872 (5.5%) | 2,490 (5.7%) | 34,763 (11.3%) | 11,686 (11.3%) | 58,729 (10.7%) | 18,668 (10.6%) | 0.00 |
| Hypoglycemia; n (%) | 4,301 (3.7%) | 1,080 (3.6%) | 4,669 (3.7%) | 1,322 (3.1%) | 11,714 (3.8%) | 4,268 (4.1%) | 20,684 (3.8%) | 6,670 (3.8%) | 0.00 |
| Hyperglycemia; n (%) | 6,940 (5.9%) | 1,796 (6.0%) | 4,682 (3.8%) | 1,805 (4.2%) | 20,768 (6.8%) | 7,619 (7.3%) | 32,390 (5.9%) | 11,220 (6.3%) | -0.02 |
| 78-07 7 7 | .,, | , , | ,, | ,, | .,, | , , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , , | |
| Disorders of fluid electrolyte and acid-base balance; n (%) | 16,879 (14.3%) | 4,101 (13.8%) | 12,788 (10.3%) | 3,971 (9.2%) | 51,918 (16.9%) | 17,299 (16.7%) | 81,585 (14.9%) | 25,371 (14.4%) | 0.01 |
| Diabetic ketoacidosis; n (%) | 8 (0.0%) | 4 (0.0%) | 4 (0.0%) | 6 (0.0%) | 59 (0.0%) | 29 (0.0%) | 071 (0.0%) | 39 (0.0%) | #DIV/0! |
| Hyperosmolar hyperglycemic nonketotic syndrome | | | | | | | | | |
| (HONK); n (%) | 735 (0.6%) | 186 (0.6%) | 558 (0.4%) | 219 (0.5%) | 1,883 (0.6%) | 782 (0.8%) | 3,176 (0.6%) | 1,187 (0.7%) | -0.01 |
| Diabetes with peripheral circulatory disorders with ICD-<br>10; n (%) | 10,913 (9.3%) | 2,930 (9.8%) | 6,325 (5.1%) | 2,235 (5.2%) | 30,630 (10.0%) | 11,331 (10.9%) | 47,868 (8.7%) | 16,496 (9.3%) | -0.02 |
| Diabetic Foot; n (%) | 4,737 (4.0%) | 1,128 (3.8%) | 4,679 (3.8%) | 1,315 (3.0%) | 14,480 (4.7%) | 4,711 (4.5%) | 23,896 (4.4%) | 7,154 (4.0%) | 0.02 |
| Gangrene ; n (%) | 897 (0.8%) | 213 (0.7%) | 1,024 (0.8%) | 259 (0.6%) | 2,075 (0.7%) | 645 (0.6%) | 3,996 (0.7%) | 1117 (0.6%) | 0.01 |
| Lower extremity amputation; n (%) | 2,269 (1.9%) | 560 (1.9%) | 1,606 (1.3%) | 406 (0.9%) | 5,709 (1.9%) | 1,731 (1.7%) | 9,584 (1.7%) | 2,697 (1.5%) | 0.02 |
| Osteomyelitis; n (%) | 1,650 (1.4%) | 400 (1.3%) | 1,708 (1.4%) | 464 (1.1%) | 3,949 (1.3%) | 1,281 (1.2%) | 7,307 (1.3%) | 2,145 (1.2%) | 0.01 |
| Skin infections; n (%) | 9,367 (8.0%) | 2,364 (7.9%) | 9,934 (8.0%) | 3,078 (7.1%) | 29,857 (9.7%) | 10,257 (9.9%) | 49,158 (9.0%) | 15,699 (8.9%) | 0.00 |
| Erectile dysfunction; n (%) | 2,941 (2.5%) | 803 (2.7%) | 2,179 (1.7%) | 898 (2.1%) | 6,731 (2.2%) | 2,409 (2.3%) | 11,851 (2.2%) | 4,110 (2.3%) | -0.01 |
| Diabetes with unspecified complication; n (%) | 6,237 (5.3%) | 1,854 (6.2%) | 4,515 (3.6%) | 1,863 (4.3%) | 16,358 (5.3%) | 6,490 (6.3%) | 27,110 (4.9%) | 10,207 (5.8%) | -0.04 |
| Diabetes mellitus without mention of complications; n | | | | | | | | | |
| (%) | 108,490 (92.2%) | 27,552 (92.6%) | 118,114 (94.8%) | 41,128 (95.0%) | 291,495 (95.2%) | 98,958 (95.4%) | 518,099 (94.4%) | 167,638 (94.8%) | -0.02 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 104,710 (89.0%) | 26,803 (90.1%) | 89,084 (71.5%) | 31,959 (73.8%) | 289,155 (94.4%) | 98,398 (94.9%) | 482,949 (88.0%) | 157,160 (88.9%) | -0.03 |
| Hyperlipidemia ; n (%) | 88,208 (75.0%) | 23,829 (80.1%) | 66,037 (53.0%) | 26,210 (60.5%) | 241,943 (79.0%) | 85,290 (82.3%) | 396,188 (72.2%) | 135,329 (76.6%) | -0.10 |
| Edema; n (%) | 12,166 (10.3%) | 3,160 (10.6%) | 8,422 (6.8%) | 2,900 (6.7%) | 43,638 (14.2%) | 15,275 (14.7%) | 64,226 (11.7%) | 21,335 (12.1%) | -0.01 |
| Renal Dysfunction (non-diabetic) ; n (%) | 34,556 (29.4%) | 8,697 (29.2%) | 24,149 (19.4%) | 7,618 (17.6%) | 101,983 (33.3%) | 33,219 (32.0%) | 160,688 (29.3%) | 49,534 (28.0%) | 0.03 |
| Occurrence of acute renal disease; n (%) | 9,176 (7.8%) | 2,303 (7.7%) | 7,529 (6.0%) | 2,364 (5.5%) | 27,683 (9.0%) | 9,014 (8.7%) | 44,388 (8.1%) | 13,681 (7.7%) | 0.01 |
| Occurrence of chronic renal insufficiency; n (%) | 26,299 (22.3%) | 6,629 (22.3%) | 15,567 (12.5%) | 4,810 (11.1%) | 80,327 (26.2%) | 25,599 (24.7%) | 122,193 (22.3%) | 37,038 (21.0%) | 0.03 |
| Chronic kidney disease ; n (%) | 25,427 (21.6%) | 6,414 (21.6%) | 15,096 (12.1%) | 4,651 (10.7%) | 76,724 (25.0%) | 24,322 (23.5%) | 117,247 (21.4%) | 35,387 (20.0%) | 0.03 |
| CKD Stage 3-4; n (%) | 16,485 (14.0%) | 4,165 (14.0%) | 9,049 (7.3%) | 2,907 (6.7%) | 50,577 (16.5%) | 15,911 (15.3%) | 76,111 (13.9%) | 22,983 (13.0%) | 0.03 |
| Occurrence of hypertensive nephropathy; n (%) | 13,898 (11.8%) | 3,469 (11.7%) | 7,405 (5.9%) | 2,248 (5.2%) | 44,203 (14.4%) | 13,558 (13.1%) | 65,506 (11.9%) | 19,275 (10.9%) | 0.03 |
| Occurrence of miscellaneous renal insufficiency; n (%) | 11,417 (9.7%) | 2,848 (9.6%) | 8,521 (6.8%) | 2,733 (6.3%) | 36,288 (11.8%) | 12,083 (11.7%) | 56,226 (10.2%) | 17,664 (10.0%) | 0.01 |
| Glaucoma or cataracts ; n (%) | 22,045 (18.7%) | 6,100 (20.5%) | 19,768 (15.9%) | 7,152 (16.5%) | 75,520 (24.7%) | 28,078 (27.1%) | 117,333 (21.4%) | 41,330 (23.4%) | -0.05 |
| Cellulitis or abscess of toe; n (%) | 2,530 (2.1%) | 580 (1.9%) | 1,977 (1.6%) | 612 (1.4%) | 6,701 (2.2%) | 2,284 (2.2%) | 11,208 (2.0%) | 3,476 (2.0%) | 0.00 |
| Foot ulcer; n (%) | 4,764 (4.0%) | 1,126 (3.8%) | 4,802 (3.9%) | 1,346 (3.1%) | 14,632 (4.8%) | 4,749 (4.6%) | 24,198 (4.4%) | 7,221 (4.1%) | 0.01 |
| Bladder stones; n (%) | 222 (0.2%) | 47 (0.2%) | 201 (0.2%) | 57 (0.1%) | 754 (0.2%) | 262 (0.3%) | 1,177 (0.2%) | 366 (0.2%) | 0.00 |
| Kidney stones; n (%) | 3,129 (2.7%) | 875 (2.9%) | 3,063 (2.5%) | 1,111 (2.6%) | 10,287 (3.4%) | 3,806 (3.7%) | 16,479 (3.0%) | 5,792 (3.3%) | -0.02 |
| Urinary tract infections (UTIs); n (%) | 15,015 (12.8%) | 3,954 (13.3%) | 11,397 (9.1%) | 3,910 (9.0%) | 58,284 (19.0%) | 22,343 (21.6%) | 84,696 (15.4%) | 30,207 (17.1%) | -0.05 |
| Dipstick urinalysis; n (%) | 41,828 (35.5%) | 12,029 (40.4%) | 36,355 (29.2%) | 14,111 (32.6%) | 136,259 (44.5%) | 50,061 (48.3%) | 214,442 (39.1%) | 76,201 (43.1%) | -0.08 |
| Non-dipstick urinalysis; n (%) | 36,680 (31.2%)<br>3,685 (3.1%) | 10,741 (36.1%)<br>966 (3.2%) | 24,847 (19.9%)<br>4,130 (3.3%) | 10,552 (24.4%)<br>1,563 (3.6%) | 99,581 (32.5%)<br>13,705 (4.5%) | 36,845 (35.5%)<br>5,353 (5.2%) | 161,108 (29.4%)<br>21,520 (3.9%) | 58,138 (32.9%)<br>7,882 (4.5%) | -0.08<br>-0.03 |
| Urine function test; n (%) Cytology; n (%) | 2,085 (1.8%) | 508 (1.7%) | 2,891 (2.3%) | 1,038 (2.4%) | 6,823 (2.2%) | 2,478 (2.4%) | 21,520 (3.9%)<br>11,799 (2.2%) | 4,024 (2.3%) | -0.03 |
| Cystos; n (%) | 2,560 (2.2%) | 656 (2.2%) | 3,232 (2.6%) | 1,103 (2.5%) | 8,994 (2.9%) | 3,007 (2.9%) | 14,786 (2.7%) | 4,766 (2.7%) | 0.00 |
| Other Covariates | -, () | | 0,202 (2.07.) | _,, | 2,00 (2.07-) | -, (=,-) | = 1,1 = 2 (= 1.1.1.) | ., (=, | |
| Liver disease; n (%) | 5,430 (4.6%) | 1,451 (4.9%) | 4,661 (3.7%) | 1,750 (4.0%) | 14,982 (4.9%) | 5,840 (5.6%) | 25,073 (4.6%) | 9,041 (5.1%) | -0.02 |
| Osteoarthritis; n (%) | 21,010 (17.9%) | 5,685 (19.1%) | 16,332 (13.1%) | 5,835 (13.5%) | 81,257 (26.5%) | 30,002 (28.9%) | 118,599 (21.6%) | 41,522 (23.5%) | -0.05 |
| Other arthritis, arthropathies and musculoskeletal pain; n | | | | | | | | | |
| (%) | 49,144 (41.8%) | 13,202 (44.4%) | 45,060 (36.2%) | 16,081 (37.1%) | 161,043 (52.6%) | 58,296 (56.2%) | 255,247 (46.5%) | 87,579 (49.6%) | -0.06 |
| Dorsopathies; n (%) | 27,972 (23.8%) | 7,679 (25.8%) | 24,944 (20.0%) | 9,217 (21.3%) | 93,330 (30.5%) | 33,983 (32.8%) | 146,246 (26.7%) | 50,879 (28.8%) | -0.05 |
| Fractures; n (%) | 5,255 (4.5%) | 1,326 (4.5%) | 5,354 (4.3%)<br>1,959 (1.6%) | 1,717 (4.0%)<br>682 (1.6%) | 18,468 (6.0%) | 6,509 (6.3%) | 29,077 (5.3%) | 9,552 (5.4%) | 0.00<br>-0.01 |
| Falls ; n (%) Osteoporosis; n (%) | 6,284 (5.3%)<br>6,103 (5.2%) | 1,678 (5.6%)<br>1,964 (6.6%) | 4,918 (3.9%) | 1,875 (4.3%) | 23,069 (7.5%)<br>24,889 (8.1%) | 8,086 (7.8%)<br>11,921 (11.5%) | 31,312 (5.7%)<br>35,910 (6.5%) | 10,446 (5.9%)<br>15,760 (8.9%) | -0.01 |
| Hyperthyroidism; n (%) | 847 (0.7%) | 274 (0.9%) | 612 (0.5%) | 277 (0.6%) | 3,328 (1.1%) | 1,334 (1.3%) | 4,787 (0.9%) | 1,885 (1.1%) | -0.03 |
| Hypothyroidism; n (%) | 17,253 (14.7%) | 5,020 (16.9%) | 11,089 (8.9%) | 4,678 (10.8%) | 50,836 (16.6%) | 19,054 (18.4%) | 79,178 (14.4%) | 28,752 (16.3%) | -0.05 |
| Other disorders of thyroid gland ; n (%) | 3,725 (3.2%) | 1,301 (4.4%) | 3,046 (2.4%) | 1,586 (3.7%) | 12,920 (4.2%) | 5,825 (5.6%) | 19,691 (3.6%) | 8,712 (4.9%) | -0.06 |
| Depression; n (%) | 12,117 (10.3%) | 3,389 (11.4%) | 9,066 (7.3%) | 3,262 (7.5%) | 44,576 (14.6%) | 16,859 (16.3%) | 65,759 (12.0%) | 23,510 (13.3%) | -0.04 |
| Anxiety; n (%) | 9,087 (7.7%) | 2,673 (9.0%) | 5,448 (4.4%) | 2,120 (4.9%) | 34,453 (11.2%) | 12,747 (12.3%) | 48,988 (8.9%) | 17,540 (9.9%) | -0.03 |
| Sleep_Disorder; n (%) | 11,137 (9.5%) | 3,176 (10.7%) | 12,982 (10.4%) | 5,001 (11.5%) | 33,719 (11.0%) | 11,667 (11.3%) | 57,838 (10.5%) | 19,844 (11.2%) | -0.02 |
| Dementia; n (%) | 8,913 (7.6%) | 2,271 (7.6%) | 6,575 (5.3%) | 1,940 (4.5%) | 39,772 (13.0%) | 14,957 (14.4%) | 55,260 (10.1%) | 19,168 (10.8%) | -0.02 |
| Delirium; n (%) | 3,536 (3.0%) | 915 (3.1%) | 3,307 (2.7%) | 1,004 (2.3%) | 13,751 (4.5%) | 5,106 (4.9%) | 20,594 (3.8%) | 7,025 (4.0%) | -0.01 |
| Psychosis; n (%) | 2,382 (2.0%) | 617 (2.1%) | 2,097 (1.7%) | 598 (1.4%) | 11,025 (3.6%) | 3,967 (3.8%) | 15,504 (2.8%) | 5,182 (2.9%) | -0.01 |
| Obesity; n (%) | 18,267 (15.5%) | 5,260 (17.7%) | 11,002 (8.8%) | 4,542 (10.5%) | 45,865 (15.0%) | 16,121 (15.5%) | 75,134 (13.7%) | 25,923 (14.7%) | -0.03<br>-0.02 |
| Overweight; n (%) | 4,108 (3.5%) | 1,280 (4.3%) | 1,273 (1.0%) | 626 (1.4%) | 10,394 (3.4%) | 3,782 (3.6%) | 15,775 (2.9%) | 5,688 (3.2%) | -0.02 |

| Smoking; n (%) | 18,795 (16.0%) | 4,685 (15.7%) | 9,206 (7.4%) | 3,169 (7.3%) | 62,562 (20.4%) | 19,676 (19.0%) | 90,563 (16.5%) | 27,530 (15.6%) | 0.02 |
|---|---|---|---|---|---|---|---|---|---|
| Alcohol abuse or dependence; n (%) | 1,421 (1.2%) | 287 (1.0%) | 966 (0.8%) | 270 (0.6%) | 2,989 (1.0%) | 901 (0.9%) | 5,376 (1.0%) | 1,458 (0.8%) | 0.02 |
| Drug abuse or dependence; n (%) | 1,825 (1.6%) | 474 (1.6%) | 875 (0.7%) | 264 (0.6%) | 4,320 (1.4%) | 1,453 (1.4%) | 7,020 (1.3%) | 2,191 (1.2%) | 0.01 |
| COPD; n (%) | 19,735 (16.8%) | 4,681 (15.7%) | 15,832 (12.7%) | 4,907 (11.3%) | 61,237 (20.0%) | 20,088 (19.4%) | 96,804 (17.6%) | 29,676 (16.8%) | 0.02 |
| Asthma; n (%) | 7,433 (6.3%) | 2,141 (7.2%) | 6,080 (4.9%) | 2,268 (5.2%) | 23,366 (7.6%) | 8,761 (8.5%) | 36,879 (6.7%) | 13,170 (7.5%) | -0.03 |
| Obstructive sleep apnea; n (%) | 10,664 (9.1%) | 3,106 (10.4%) | 10,321 (8.3%) | 4,281 (9.9%) | 26,855 (8.8%) | 9,150 (8.8%) | 47,840 (8.7%) | 16,537 (9.4%) | -0.02 |
| Pneumonia; n (%) | 7,668 (6.5%) | 1,657 (5.6%) | 7,710 (6.2%) | 2,240 (5.2%) | 23,525 (7.7%) | 7,763 (7.5%) | 38,903 (7.1%) | 11,660 (6.6%) | 0.02 |
| Imaging; n (%) | 634 (0.5%) | 128 (0.4%) | 394 (0.3%) | 119 (0.3%) | 1,614 (0.5%) | 554 (0.5%) | 2,642 (0.5%) | 801 (0.5%) | 0.00 |
| Diabetes Medications | | | | | | | | | |
| DM Medications - AGIs; n (%) | 372 (0.3%) | 96 (0.3%) | 376 (0.3%) | 139 (0.3%) | 1,037 (0.3%) | 431 (0.4%) | 1,785 (0.3%) | 666 (0.4%) | -0.02 |
| DM Medications - Glitazones; n (%) | 8,229 (7.0%) | 2,709 (9.1%) | 10,908 (8.8%) | 4,523 (10.4%) | 12,093 (3.9%) | 6,087 (5.9%) | 31,230 (5.7%) | 13,319 (7.5%) | -0.07 |
| DM Medications - GLP-1 RA; n (%) | 509 (0.4%) | 191 (0.6%) | 563 (0.5%) | 188 (0.4%) | 850 (0.3%) | 342 (0.3%) | 1,922 (0.4%) | #VALUE! | #VALUE! |
| DM Medications - Insulin; n (%) | 15,960 (13.6%) | 5,836 (19.6%) | 15,477 (12.4%) | 6,702 (15.5%) | 49,256 (16.1%) | 22,937 (22.1%) | 80,693 (14.7%) | 35,475 (20.1%) | -0.14 |
| DM Medications - Meglitinides; n (%) | 942 (0.8%) | 677 (2.3%) | 1,640 (1.3%) | 1,574 (3.6%) | 3,540 (1.2%) | 3,201 (3.1%) | 6,122 (1.1%) | 5,452 (3.1%) | -0.14 |
| DM Medications - Metformin; n (%) | 56,560 (48.1%) | 17,047 (57.3%) | 58,461 (46.9%) | 25,481 (58.8%) | 135,361 (44.2%) | 57,121 (55.1%) | 250,382 (45.6%) | 99,649 (56.4%) | -0.22 |
| Concomitant initiation or current use of SGLT2i; n (%) | 994 (0.8%) | 436 (1.5%) | 690 (0.6%) | 575 (1.3%) | 1,805 (0.6%) | 1,291 (1.2%) | 3,489 (0.6%) | 2,302 (1.3%) | -0.07 |
| Concomitant initiation or current use of AGIs; n (%) | 253 (0.2%) | 64 (0.2%) | 280 (0.2%) | 92 (0.2%) | 704 (0.2%) | 304 (0.3%) | 1,237 (0.2%) | 460 (0.3%) | -0.02 |
| Concomitant initiation or current use of Glitazones; n (%) | 5,587 (4.7%) | 1,440 (4.8%) | 7,210 (5.8%) | 2,282 (5.3%) | 7,638 (2.5%) | 3,431 (3.3%) | 20,435 (3.7%) | 7,153 (4.0%) | -0.02 |
| 6 | 227 (2.20() | 50 (0.20() | 242 (0.20() | 57 (0.40() | 227 (2.40() | 442 (0.40() | (0.44.1151 | (0.441.15) | 10.441.1151 |
| Concomitant initiation or current use of GLP-1 RA; n (%) | 227 (0.2%) | 68 (0.2%) | 312 (0.3%) | 57 (0.1%) | 327 (0.1%) | 113 (0.1%) | #VALUE! | #VALUE! | #VALUE! |
| C | 10,116 (8.6%) | 3,986 (13.4%) | 9,739 (7.8%) | 4,333 (10.0%) | 31,424 (10.3%) | 15,966 (15.4%) | 51,279 (9.3%) | 24,285 (13.7%) | -0.14 |
| Concomitant initiation or current use of Insulin; n (%) Concomitant initiation or current use of Meglitinides; n | 10,116 (8.6%) | 3,986 (13.4%) | 9,739 (7.8%) | 4,333 (10.0%) | 31,424 (10.3%) | 15,966 (15.4%) | 51,279 (9.3%) | 24,285 (13.7%) | -0.14 |
| (%) | 535 (0.5%) | 485 (1.6%) | 950 (0.8%) | 1,104 (2.5%) | 2,171 (0.7%) | 2,367 (2.3%) | 3,656 (0.7%) | 3,956 (2.2%) | -0.13 |
| (76) | 333 (0.3%) | 463 (1.0%) | 330 (0.8%) | 1,104 (2.570) | 2,171 (0.776) | 2,307 (2.370) | 3,030 (0.778) | 3,530 (2.270) | -0.13 |
| Concomitant initiation or current use of Metformin; n (%) | 42,837 (36.4%) | 13,655 (45.9%) | 44,541 (35.7%) | 20,708 (47.8%) | 98,310 (32.1%) | 44,919 (43.3%) | 185,688 (33.8%) | 79,282 (44.9%) | -0.23 |
| Past use of SGLT2i; n (%) | 445 (0.4%) | 209 (0.7%) | 315 (0.3%) | 214 (0.5%) | 1,055 (0.3%) | 568 (0.5%) | 1,815 (0.3%) | 991 (0.6%) | -0.04 |
| Past use of AGIs ; n (%) | 119 (0.1%) | 32 (0.1%) | 96 (0.1%) | 47 (0.1%) | 333 (0.1%) | 127 (0.1%) | 548 (0.1%) | 206 (0.1%) | 0.00 |
| | | | | | | | | | -0.09 |
| Past use of Glitazones ; n (%) | 2,642 (2.2%) | 1,269 (4.3%) | 3,699 (3.0%) | 2,241 (5.2%) | 4,455 (1.5%) | 2,656 (2.6%) | 10,796 (2.0%) | 6,166 (3.5%) | -0.09 |
| Past use of GLP-1 RA; n (%) | 292 (0.2%) | 124 (0.4%) | 255 (0.2%) | 134 (0.3%) | 523 (0.2%) | 229 (0.2%) | 1,070 (0.2%) | 487 (0.3%) | |
| Past use of Insulin ; n (%) | 5,844 (5.0%) | 1,850 (6.2%) | 5,738 (4.6%) | 2,370 (5.5%) | 17,835 (5.8%) | 6,974 (6.7%) | 29,417 (5.4%) | 11,194 (6.3%) | -0.04 |
| Past use of Meglitinides ; n (%) | 407 (0.3%) | 192 (0.6%) | 690 (0.6%) | 470 (1.1%) | 1,369 (0.4%) | 834 (0.8%) | 2,466 (0.4%) | 1,496 (0.8%) | -0.05 |
| Past use of metformin (final); n (%) | 13,723 (11.7%) | 3,392 (11.4%) | 13,920 (11.2%) | 4,773 (11.0%) | 37,051 (12.1%) | 12,202 (11.8%) | 64,694 (11.8%) | 20,367 (11.5%) | 0.01 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 54,239 (46.1%) | 12,202 (41.0%) | 56,542 (45.4%) | 18,022 (41.6%) | 131,273 (42.9%) | 40,555 (39.1%) | 242,054 (44.1%) | 70,779 (40.0%) | 0.08 |
| Use of ARBs; n (%) | 25,030 (21.3%) | 8,315 (27.9%) | 28,565 (22.9%) | 12,351 (28.5%) | 76,768 (25.1%) | 32,742 (31.6%) | 130,363 (23.8%) | 53,408 (30.2%) | -0.14 |
| Use of Loop Diuretics - ; n (%) | 28,952 (24.6%) | 6,708 (22.5%) | 30,314 (24.3%) | 9,013 (20.8%) | 93,126 (30.4%) | 29,520 (28.5%) | 152,392 (27.8%) | 45,241 (25.6%) | 0.05 |
| Use of other diuretics-; n (%) | 5,674 (4.8%) | 1,464 (4.9%) | 6,178 (5.0%) | 2,066 (4.8%) | 17,047 (5.6%) | 5,658 (5.5%) | 28,899 (5.3%) | 9,188 (5.2%) | 0.00 |
| Use of nitrates-; n (%) | 17,689 (15.0%) | 4,233 (14.2%) | 21,232 (17.0%) | 6,834 (15.8%) | 52,053 (17.0%) | 17,114 (16.5%) | 90,974 (16.6%) | 28,181 (15.9%) | 0.02 |
| Use of other hypertension drugs; n (%) | 12,758 (10.8%) | 2,776 (9.3%) | 12,657 (10.2%) | 3,485 (8.0%) | 37,331 (12.2%) | 11,366 (11.0%) | 62,746 (11.4%) | 17,627 (10.0%) | 0.05 |
| Use of digoxin-; n (%) | 5,809 (4.9%) | 1,265 (4.3%) | 7,057 (5.7%) | 2,115 (4.9%) | 17,623 (5.8%) | 5,746 (5.5%) | 30,489 (5.6%) | 9,126 (5.2%) | 0.02 |
| Use of Anti-arrhythmics; n (%) | 4,023 (3.4%) | 1,037 (3.5%) | 5,048 (4.1%) | 1,661 (3.8%) | 13,423 (4.4%) | 4,451 (4.3%) | 22,494 (4.1%) | 7,149 (4.0%) | 0.01 |
| Use of COPD/asthma meds-; n (%) | 18,132 (15.4%) | 5,349 (18.0%) | 20,060 (16.1%) | 7,587 (17.5%) | 57,441 (18.8%) | 22,852 (22.0%) | 95,633 (17.4%) | 35,788 (20.2%) | -0.07 |
| Use of statins; n (%) | 78,990 (67.1%) | 21,287 (71.5%) | 84,053 (67.5%) | 31,003 (71.6%) | 212,184 (69.3%) | 75,861 (73.2%) | 375,227 (68.4%) | 128,151 (72.5%) | -0.09 |
| Use of other lipid-lowering drugs; n (%) | 14,917 (12.7%) | 4,648 (15.6%) | 20,396 (16.4%) | 8,393 (19.4%) | 36,070 (11.8%) | 14,623 (14.1%) | 71,383 (13.0%) | 27,664 (15.7%) | -0.08 |
| Use of antiplatelet agents; n (%) | 32,387 (27.5%) | 8,801 (29.6%) | 40,482 (32.5%) | 14,677 (33.9%) | 84,313 (27.5%) | 30,711 (29.6%) | 157,182 (28.7%) | 54,189 (30.7%) | -0.04 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | | | | | | | | | |
| Apixaban, Warfarin); n (%) | 13,819 (11.7%) | 3,377 (11.3%) | 15,147 (12.2%) | 4,720 (10.9%) | 48,289 (15.8%) | 15,695 (15.1%) | 77,255 (14.1%) | 23,792 (13.5%) | 0.02 |
| Use of heparin and other low-molecular weight heparins; | | | | | | | | | |
| n (%) | 1,120 (1.0%) | 249 (0.8%) | 84 (0.1%) | 31 (0.1%) | 2,943 (1.0%) | 937 (0.9%) | 4,147 (0.8%) | 1,217 (0.7%) | 0.01 |
| Use of NSAIDs; n (%) | 14,354 (12.2%) | 4,038 (13.6%) | 15,019 (12.1%) | 5,782 (13.4%) | 42,896 (14.0%) | 17,195 (16.6%) | 72,269 (13.2%) | 27,015 (15.3%) | -0.06 |
| Use of oral corticosteroids; n (%) | 20,557 (17.5%) | 5,245 (17.6%) | 21,988 (17.6%) | 7,546 (17.4%) | 66,685 (21.8%) | 22,585 (21.8%) | 109,230 (19.9%) | 35,376 (20.0%) | 0.00 |
| Use of bisphosphonate (); n (%) | 2,897 (2.5%) | 926 (3.1%) | 3,145 (2.5%) | 1,139 (2.6%) | 9,018 (2.9%) | 4,530 (4.4%) | 15,060 (2.7%) | 6,595 (3.7%) | -0.06 |
| Use of opioids-; n (%) | 35,963 (30.6%) | 9,123 (30.7%) | 40,525 (32.5%) | 13,385 (30.9%) | 100,549 (32.8%) | 33,144 (32.0%) | 177,037 (32.3%) | 55,652 (31.5%) | 0.02 |
| Use of antidepressants; n (%) | 27,916 (23.7%) | 7,888 (26.5%) | 28,755 (23.1%) | 10,402 (24.0%) | 86,397 (28.2%) | 32,027 (30.9%) | 143,068 (26.1%) | 50,317 (28.5%) | -0.05 |
| Use of antipsychotics; n (%) | 3,309 (2.8%) | 989 (3.3%) | 3,200 (2.6%) | 1,004 (2.3%) | 13,359 (4.4%) | 5,613 (5.4%) | 19,868 (3.6%) | 7,606 (4.3%) | -0.04 |
| Use of anticonvulsants; n (%) | 19,086 (16.2%) | 5,320 (17.9%) | 17,058 (13.7%) | 6,022 (13.9%) | 62,576 (20.4%) | 22,838 (22.0%) | 98,720 (18.0%) | 34,180 (19.3%) | -0.03 |
| Use of lithium-; n (%) | 152 (0.1%) | 46 (0.2%) | 176 (0.1%) | 63 (0.1%) | 380 (0.1%) | 124 (0.1%) | 708 (0.1%) | 233 (0.1%) | 0.00 |
| Use of Benzos-; n (%) | 11,453 (9.7%) | 3,378 (11.4%) | 17,055 (13.7%) | 5,882 (13.6%) | 37,412 (12.2%) | 13,247 (12.8%) | 65,920 (12.0%) | 22,507 (12.7%) | -0.02 |
| Use of anxiolytics/hypnotics-; n (%) | 7,983 (6.8%) | 2,254 (7.6%) | 9,769 (7.8%) | 3,688 (8.5%) | 22,911 (7.5%) | 9,271 (8.9%) | 40,663 (7.4%) | 15,213 (8.6%) | -0.04 |
| Use of dementia meds-; n (%) | 4,036 (3.4%) | 1,145 (3.8%) | 4,105 (3.3%) | 1,213 (2.8%) | 20,223 (6.6%) | 8,743 (8.4%) | 28,364 (5.2%) | 11,101 (6.3%) | -0.05 |
| Use of antiparkinsonian meds-; n (%) | 3,220 (2.7%) | 916 (3.1%) | 3,571 (2.9%) | 1,193 (2.8%) | 12,914 (4.2%) | 4,733 (4.6%) | 19,705 (3.6%) | 6,842 (3.9%) | -0.02 |
| Any use of pramlintide; n (%) | 17 (0.0%) | 9 (0.0%) | 49 (0.0%) | 37 (0.1%) | 24 (0.0%) | 29 (0.0%) | 090 (0.0%) | 075 (0.0%) | #DIV/0! |
| Any use of 1st generation sulfonylureas; n (%) | 80 (0.1%) | 11 (0.0%) | 190 (0.2%) | 15 (0.0%) | 210 (0.1%) | 27 (0.0%) | 480 (0.1%) | 053 (0.0%) | 0.00 |
| Entresto (sacubitril/valsartan); n (%) | 189 (0.2%) | 65 (0.2%) | 44 (0.0%) | 20 (0.0%) | 248 (0.1%) | 120 (0.1%) | 481 (0.1%) | 205 (0.1%) | 0.00 |
| · | / | / | 1 / | / | - (- /-/ | / | - 1 / | | |

| Initiation as monotherapy v4 ; n (%) | 30,107 (25.6%) | 7,242 (24.3%) | 29,945 (24.0%) | 10,416 (24.1%) | 63,712 (20.8%) | 20,833 (20.1%) | 123,764 (22.6%) | 38,491 (21.8%) | 0.02 |
|---|---|---|---|---|---|---|---|---|---|
| Labs | | | | | | | 242,279 | 73,065 | |
| Lab values- HbA1c (%); n (%) | 29,636 (25.2%) | 8,836 (29.7%) | 4,979 (4.0%) | 1,899 (4.4%) | N/A | N/A | 34,615 (14.3%) | 10,735 (14.7%) | -0.01 |
| Lab values- HbA1c (%) (within 3 months); n (%) | 22,154 (18.8%) | 6,713 (22.6%) | 3,792 (3.0%) | 1,466 (3.4%) | N/A | N/A | 25,946 (10.7%) | 8,179 (11.2%) | -0.02 |
| Lab values- HbA1c (%) (within 6 months); n (%) | 29,636 (25.2%) | 8,836 (29.7%) | 4,979 (4.0%) | 1,899 (4.4%) | N/A | N/A | 34,615 (14.3%) | 10,735 (14.7%) | -0.01 |
| Lab values- BNP; n (%) | 1,183 (1.0%) | 355 (1.2%) | 168 (0.1%) | 74 (0.2%) | N/A | N/A | 1,351 (0.6%) | 429 (0.6%) | 0.00 |
| Lab values- BNP (within 3 months); n (%) | 761 (0.6%) | 220 (0.7%) | 112 (0.1%) | 54 (0.1%) | N/A | N/A | 873 (0.4%) | 274 (0.4%) | 0.00 |
| Lab values-BNP (within 6 months); n (%) | 1,183 (1.0%) | 355 (1.2%) | 168 (0.1%) | 74 (0.2%) | N/A | N/A | 1,351 (0.6%) | 429 (0.6%) | 0.00 |
| Lab values- BUN (mg/dl); n (%) | 32,750 (27.8%) | 9,782 (32.9%) | 4,699 (3.8%) | 2,083 (4.8%) | N/A | N/A | 37,449 (15.5%) | 11,865 (16.2%) | -0.02 |
| , , , , | | | | | | N/A | | | -0.02 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 24,568 (20.9%) | 7,492 (25.2%) | 3,526 (2.8%) | 1,589 (3.7%) | N/A | • | 28,094 (11.6%) | 9,081 (12.4%) | |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 32,750 (27.8%) | 9,782 (32.9%) | 4,699 (3.8%) | 2,083 (4.8%) | N/A | N/A | 37,449 (15.5%) | 11,865 (16.2%) | -0.02 |
| Lab values- Creatinine (mg/dl) ; n (%) | 33,612 (28.6%) | 10,026 (33.7%) | 4,992 (4.0%) | 2,214 (5.1%) | N/A | N/A | 38,604 (15.9%) | 12,240 (16.8%) | -0.02 |
| Lab values- Creatinine (mg/dl) (within 3 months); n (%) | 25,223 (21.4%) | 7,691 (25.8%) | 3,751 (3.0%) | 1,680 (3.9%) | N/A | N/A | 28,974 (12.0%) | 9,371 (12.8%) | -0.02 |
| Lab values- Creatinine (mg/dl) (within 6 months); n (%) | 33,612 (28.6%) | 10,026 (33.7%) | 4,992 (4.0%) | 2,214 (5.1%) | N/A | N/A | 38,604 (15.9%) | 12,240 (16.8%) | -0.02 |
| Lab values- HDL level (mg/dl); n (%) | 25,367 (21.6%) | 7,868 (26.4%) | 4,371 (3.5%) | 1,733 (4.0%) | N/A | N/A | 29,738 (12.3%) | 9,601 (13.1%) | -0.02 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 17,842 (15.2%) | 5,652 (19.0%) | 3,126 (2.5%) | 1,273 (2.9%) | N/A | N/A | 20,968 (8.7%) | 6,925 (9.5%) | -0.03 |
| Lab values- FIDE level (Hig/ul) (within 5 months), ii (%) | 17,642 (13.2%) | 3,032 (19.0%) | 3,120 (2.3%) | 1,273 (2.9%) | N/A | N/A | 20,900 (6.7%) | 0,923 (9.5%) | -0.03 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 25,367 (21.6%) | 7,868 (26.4%) | 4,371 (3.5%) | 1,733 (4.0%) | N/A | N/A | 29,738 (12.3%) | 9,601 (13.1%) | -0.02 |
| Lab values- LDL level (mg/dl); n (%) | 26,132 (22.2%) | 8,058 (27.1%) | 4,734 (3.8%) | 1,843 (4.3%) | N/A | N/A | 30,866 (12.7%) | 9,901 (13.6%) | -0.03 |
| 3, 1, | -, - , - , | -,, | , . ( , | , ( , | • | • | , , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | |
| Lab values- LDL level (mg/dl) (within 3 months); n (%) | 18,361 (15.6%) | 5,776 (19.4%) | 3,399 (2.7%) | 1,353 (3.1%) | N/A | N/A | 21,760 (9.0%) | 7,129 (9.8%) | -0.03 |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 26,132 (22.2%) | 8,058 (27.1%) | 4,734 (3.8%) | 1,843 (4.3%) | N/A | N/A | 30,866 (12.7%) | 9,901 (13.6%) | -0.03 |
| Lab values- NT-proBNP; n (%) | 147 (0.1%) | 44 (0.1%) | 13 (0.0%) | 4 (0.0%) | N/A | N/A | 160 (0.1%) | 48 (0.1%) | 0.00 |
| Lab values- NT-proBNP (within 3 months); n (%) | 87 (0.1%) | 20 (0.1%) | 7 (0.0%) | 2 (0.0%) | N/A | N/A | 94 (0.0%) | 22 (0.0%) | - |
| Lab values- NT-proBNP (within 5 months); n (%) | 147 (0.1%) | 44 (0.1%) | 13 (0.0%) | | | N/A | | 48 (0.1%) | |
| | | | | 4 (0.0%) | N/A | | 160 (0.1%) | | -0.03 |
| Lab values-Total cholesterol (mg/dl); n (%) | 25,813 (21.9%) | 7,987 (26.8%) | 4,557 (3.7%) | 1,811 (4.2%) | N/A | N/A | 30,370 (12.5%) | 9,798 (13.4%) | -0.03 |
| Lab values- Total cholesterol (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 18,137 (15.4%) | 5,731 (19.3%) | 3,255 (2.6%) | 1,323 (3.1%) | N/A | N/A | 21,392 (8.8%) | 7,054 (9.7%) | -0.03 |
| Lab values-Total cholesterol (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 25,813 (21.9%) | 7,987 (26.8%) | 4,557 (3.7%) | 1,811 (4.2%) | N/A | N/A | 30,370 (12.5%) | 9,798 (13.4%) | -0.03 |
| Lab values-Triglyceride level (mg/dl); n (%) | 25,491 (21.7%) | 7,878 (26.5%) | 4,465 (3.6%) | 1,779 (4.1%) | N/A | N/A | 29,956 (12.4%) | 9,657 (13.2%) | -0.02 |
| Lab values-Triglyceride level (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 17,919 (15.2%) | 5,649 (19.0%) | 3,196 (2.6%) | 1,307 (3.0%) | N/A | N/A | 21,115 (8.7%) | 6,956 (9.5%) | -0.03 |
| Lab values-Triglyceride level (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 25,491 (21.7%) | 7,878 (26.5%) | 4,465 (3.6%) | 1,779 (4.1%) | N/A | N/A | 29,956 (12.4%) | 9,657 (13.2%) | -0.02 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | | | | | | | | | |
| included) v4 | 29,363 | 8,750 | 4,334 | 1,833 | N/A | N/A | 33,697 | 10,583 | |
| mean (sd) | 7.89 (1.77) | 7.78 (1.69) | 8.01 (1.85) | 7.92 (1.76) | N/A | N/A | 7.91 (1.78) | 7.80 (1.70) | 0.06 |
| median [IQR] | 7.45 [6.70, 8.65] | 7.40 [6.60, 8.50] | 7.50 [6.70, 8.80] | 7.50 [6.70, 8.70] | N/A | N/A | 7.46 (1.78) | 7.42 (1.70) | 0.02 |
| Missing; n (%) | 88,322 (75.0%) | 21,009 (70.6%) | 120,260 (96.5%) | 41,473 (95.8%) | N/A | N/A | 208,582 (86.1%) | 62,482 (85.5%) | 0.02 |
| Lab result number- BNP mean | 1,183 | 355 | 168 | 74 | N/A | N/A | 1,351 | 429 | 0.02 |
| | | | | * * | | | | | 0.20 |
| mean (sd) | 302.70 (552.45) | 212.12 (352.66) | 339.91 (671.94) | 210.76 (314.60) | N/A | N/A | 307.33 (568.82) | 211.89 (346.86) | 0.20 |
| median [IQR] | 127.33 [46.80, 331.80] | 106.50 [36.60, 238.00] | 93.50 [37.50, 330.50] | 100.50 [30.75, 261.62] | N/A | N/A | #VALUE! | 105.47 (346.86) | #VALUE! |
| Missing; n (%) | 116,502 (99.0%) | 29,404 (98.8%) | 124,426 (99.9%) | 43,232 (99.8%) | N/A | N/A | 240,928 (99.4%) | 72,636 (99.4%) | 0.00 |
| Lab result number- BUN (mg/dl) mean | 32,750 | 9,782 | 4,699 | 2,083 | N/A | N/A | 37,449 | 11,865 | |
| mean (sd) | 20.84 (10.09) | 20.26 (9.38) | 705.76 (11,062.74) | 217.15 (4,979.06) | N/A | N/A | 106.78 (3918.48) | 54.83 (2085.99) | 0.02 |
| median [IQR] | 18.33 [14.50, 24.33] | 18.00 [14.00, 23.75] | 18.00 [14.00, 23.00] | 17.00 [14.00, 22.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 84,935 (72.2%) | 19,977 (67.1%) | 119,895 (96.2%) | 41,223 (95.2%) | N/A | N/A | 204,830 (84.5%) | 61,200 (83.8%) | 0.02 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 to | | | | | | | | | |
| 15 included) | 33,274 | 9,917 | 4,811 | 2,079 | N/A | N/A | 38,085 | 11,996 | |
| mean (sd) | 1.16 (0.58) | 1.13 (0.55) | 1.11 (0.58) | 1.05 (0.51) | N/A | N/A | 1.15 (0.58) | 1.12 (0.54) | 0.05 |
| median [IQR] | 1.04 [0.85, 1.31] | 1.02 [0.84, 1.28] | 1.00 [0.83, 1.22] | 0.98 [0.81, 1.15] | N/A | N/A | 1.03 (0.58) | 1.01 (0.54) | 0.04 |
| Missing; n (%) | 84,411 (71.7%) | 19,842 (66.7%) | 119,783 (96.1%) | 41,227 (95.2%) | N/A | N/A | 204,194 (84.3%) | 61,069 (83.6%) | 0.02 |
| | 04,411 (71.7%) | 19,042 (00.7%) | 119,765 (90.176) | 41,227 (93.2%) | IN/A | N/A | 204,194 (64.5%) | 01,009 (03.0%) | 0.02 |
| Lab result number- HDL level (mg/dl) mean (only =<5000 | 25.257 | 7.000 | 4.057 | 4.700 | **/* | N1/* | 20.724 | 0.000 | |
| included) | 25,367 | 7,868 | 4,357 | 1,732 | N/A | N/A | 29,724 | 9,600 | |
| mean (sd) | 44.55 (13.79) | 45.39 (14.02) | 44.51 (66.02) | 43.66 (14.21) | N/A | N/A | 44.54 (28.30) | 45.08 (14.06) | -0.02 |
| median [IQR] | 43.00 [35.50, 52.00] | 44.00 [36.00, 53.00] | 42.00 [35.00, 50.00] | 42.00 [35.00, 51.00] | N/A | N/A | 42.85 (28.30) | 43.64 (14.06) | -0.04 |
| Missing; n (%) | 92,318 (78.4%) | 21,891 (73.6%) | 120,237 (96.5%) | 41,574 (96.0%) | N/A | N/A | 212,555 (87.7%) | 63,465 (86.9%) | 0.02 |
| Lab result number- LDL level (mg/dl) mean (only =<5000 | | | | | | | | | |
| included) | 25,614 | 7,895 | 4,389 | 1,745 | N/A | N/A | 30,003 | 9,640 | |
| mean (sd) | 85.78 (41.18) | 83.18 (39.96) | 88.03 (42.48) | 86.46 (42.72) | N/A | N/A | 86.11 (41.37) | 83.77 (40.48) | 0.06 |
| median [IQR] | 82.00 [61.00, 109.00] | 79.40 [59.00, 104.00] | 85.00 [62.00, 111.00] | 83.00 [62.00, 110.50] | N/A | N/A | 82.44 (41.37) | 80.05 (40.48) | 0.06 |
| Missing; n (%) | 92,071 (78.2%) | 21,864 (73.5%) | 120,205 (96.5%) | 41,561 (96.0%) | N/A | N/A | 212,276 (87.6%) | 63,425 (86.8%) | 0.02 |
| ·· 0/ 1/1/ | , (- 3.270) | ,, | | , ( 0,0) | .,,,, | ,,,, | , (23/0) | , (0,0) | |

| Lab result number-Total cholesterol (mg/dl) mean (only | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| =<5000 included) | 25,796 | 7,976 | 4,539 | 1,807 | N/A | N/A | 30,335 | 9,783 | |
| mean (sd) | 170.43 (50.39) | 167.26 (48.36) | 173.43 (50.55) | 171.71 (52.14) | N/A | N/A | 170.88 (50.41) | 168.08 (49.08) | 0.06 |
| median [IQR] | | | | 166.00 [140.00, 198.00] | N/A | N/A | 164.45 (50.41) | 161.92 (49.08) | 0.05 |
| Missing; n (%) | 91,889 (78.1%) | 21,783 (73.2%) | 120,055 (96.4%) | 41,499 (95.8%) | N/A | N/A | 211,944 (87.5%) | 63,282 (86.6%) | 0.03 |
| Lab result number-Triglyceride level (mg/dl) mean (only | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ,, | .,, | ,, | • | • | , | , . (, | |
| =<5000 included) | 25,488 | 7,878 | 4,450 | 1,778 | N/A | N/A | 29,938 | 9,656 | |
| mean (sd) | 185.44 (156.55) | 178.86 (148.70) | 192.77 (168.94) | 192.68 (182.22) | N/A | N/A | 186.53 (158.46) | 181.40 (155.42) | 0.03 |
| median [IQR] | 150.00 [107.00, 217.00] | 146.00 [104.00, 210.00] | 152.25 [109.00, 220.62] | 150.00 [106.00, 221.00] | N/A | N/A | 150.33 (158.46) | 146.74 (155.42) | 0.02 |
| Missing; n (%) | 92,197 (78.3%) | 21,881 (73.5%) | 120,144 (96.4%) | 41,528 (95.9%) | N/A | N/A | 212,341 (87.6%) | 63,409 (86.8%) | 0.02 |
| Lab result number- Hemoglobin mean (only >0 included) | 23,872 | 7,214 | 3,292 | 1,439 | N/A | N/A | 27,164 | 8,653 | |
| mean (sd) | 13.24 (1.82) | 13.26 (1.76) | 5,116.60 (195,020.21) | 313.03 (6,066.36) | N/A | N/A | 631.72 (67884.51) | 63.11 (2473.43) | 0.01 |
| median [IQR] | 13.30 [12.05, 14.50] | 13.30 [12.10, 14.50] | 13.50 [12.20, 14.65] | 13.50 [12.25, 14.70] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 93,813 (79.7%) | 22,545 (75.8%) | 121,302 (97.4%) | 41,867 (96.7%) | N/A | N/A | 215,115 (88.8%) | 64,412 (88.2%) | 0.02 |
| Lab result number- Serum sodium mean (only > 90 and < | | | | | | | | | |
| 190 included) | 32,487 | 9,706 | 4,212 | 1,898 | N/A | N/A | 36,699 | 11,604 | |
| mean (sd) | 139.35 (2.92) | 139.52 (2.83) | 138.95 (2.86) | 139.10 (2.73) | N/A | N/A | 139.30 (2.91) | 139.45 (2.81) | -0.05 |
| median [IQR] | 139.50 [138.00, 141.00] | 140.00 [138.00, 141.33] | 139.00 [137.25, 141.00] | 139.00 [137.65, 141.00] | N/A | N/A | 139.44 (2.91) | 139.84 (2.81) | -0.14 |
| Missing; n (%) | 85,198 (72.4%) | 20,053 (67.4%) | 120,382 (96.6%) | 41,408 (95.6%) | N/A | N/A | 205,580 (84.9%) | 61,461 (84.1%) | 0.02 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | |
| included) | 29,792 | 9,021 | 3,808 | 1,707 | N/A | N/A | 33,600 | 10,728 | |
| mean (sd) | 4.16 (0.35) | 4.17 (0.35) | 4.15 (0.50) | 4.14 (0.59) | N/A | N/A | 4.16 (0.37) | 4.17 (0.40) | -0.03 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.45] | N/A | N/A | 4.20 (0.37) | 4.20 (0.40) | 0.00 |
| Missing; n (%) | 87,893 (74.7%) | 20,738 (69.7%) | 120,786 (96.9%) | 41,599 (96.1%) | N/A | N/A | 208,679 (86.1%) | 62,337 (85.3%) | 0.02 |
| Lab result number- Glucose (fasting or random) mean | | | | | | | | | |
| (only 10-1000 included) | 32,468 | 9,708 | 4,185 | 1,876 | N/A | N/A | 36,653 | 11,584 | |
| mean (sd) | 166.92 (73.20) | 161.27 (67.25) | 170.78 (75.20) | 164.77 (71.73) | N/A | N/A | 167.36 (73.43) | 161.84 (68.00) | 0.08 |
| median [IQR] | 148.00 [119.00, 193.00] | 144.00 [117.00, 185.00] | 151.00 [121.00, 198.75] | 145.00 [119.08, 189.00] | N/A | N/A | 148.34 (73.43) | 144.16 (68.00) | 0.06 |
| Missing; n (%) | 85,217 (72.4%) | 20,051 (67.4%) | 120,409 (96.6%) | 41,430 (95.7%) | N/A | N/A | 205,626 (84.9%) | 61,481 (84.1%) | 0.02 |
| Lab result number- Potassium mean (only 1-7 included) | 33,114 | 9,891 | 4,624 | 2,044 | N/A | N/A | 37,738 | 11,935 | |
| mean (sd) | 4.45 (0.46) | 4.43 (0.45) | 4.38 (0.45) | 4.38 (0.44) | N/A | N/A | 4.44 (0.46) | 4.42 (0.45) | 0.04 |
| median [IQR] | 4.40 [4.15, 4.70] | 4.40 [4.12, 4.70] | 4.40 [4.10, 4.70] | 4.40 [4.10, 4.65] | N/A | N/A | 4.40 (0.46) | 4.40 (0.45) | 0.00 |
| Missing; n (%) | 84,571 (71.9%) | 19,868 (66.8%) | 119,970 (96.3%) | 41,262 (95.3%) | N/A | N/A | 204,541 (84.4%) | 61,130 (83.7%) | 0.02 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 3.56 (2.35) | 3.54 (2.35) | 2.65 (2.17) | 2.56 (2.12) | 4.15 (2.42) | 4.19 (2.41) | 3.68 (2.35) | 3.68 (2.33) | 0.00 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 4.00 [2.00, 6.00] | 4.00 [2.00, 6.00] | 3.33 (2.35) | 3.34 (2.33) | 0.00 |
| Frailty Score: Qualitative Version 365 days as Categories, | | | | | | | | | |
| v1 | | | | | | | | | |
| 0; n (%) | 21,406 (18.2%) | 5,871 (19.7%) | 6,853 (5.5%) | 3,610 (8.3%) | 41,807 (13.6%) | 15,665 (15.1%) | 70,066 (12.8%) | 25,146 (14.2%) | -0.04 |
| 1 to 2; n (%) | 39,327 (33.4%) | 10,519 (35.3%) | 51,129 (41.0%) | 18,494 (42.7%) | 73,716 (24.1%) | 24,561 (23.7%) | 164,172 (29.9%) | 53,574 (30.3%) | -0.01 |
| 3 or more; n (%) | 56,952 (48.4%) | 13,369 (44.9%) | 66,612 (53.5%) | 21,202 (49.0%) | 190,781 (62.3%) | 63,451 (61.2%) | 314,345 (57.3%) | 98,022 (55.5%) | 0.04 |
| Frailty Score: Empirical Version 365 days as Categories, | | | | | | | | | |
| <0.12908; n (%) | 5,864 (5.0%) | 1,676 (5.6%) | 6,888 (5.5%) | 2,978 (6.9%) | 5,981 (2.0%) | 2,264 (2.2%) | 18,733 (3.4%) | 6,918 (3.9%) | -0.03 |
| 0.12908 - 0.1631167; n (%) | 24,734 (21.0%) | 6,531 (21.9%) | 27,427 (22.0%) | 10,535 (24.3%) | 31,035 (10.1%) | 10,737 (10.4%) | 83,196 (15.2%) | 27,803 (15.7%) | -0.01 |
| >= 0.1631167; n (%) | 87,087 (74.0%) | 21,552 (72.4%) | 90,279 (72.5%) | 29,793 (68.8%) | 269,288 (87.9%) | 90,676 (87.5%) | 446,654 (81.4%) | 142,021 (80.4%) | 0.03 |
| Non-Frailty; n (%) | 62,261 (52.9%) | 16,998 (57.1%) | 58,216 (46.7%) | 21,937 (50.7%) | 11,446 (3.7%) | 3,726 (3.6%) | 131,923 (24.0%) | 42,661 (24.1%) | 0.00 |
| Fully Constitution of Contract | | | | | | | | | |
| Frailty Score (mean): Qualitative Version 365 days, v1 | 2.07.(2.65) | 2.75 (2.55) | 2.40 (2.20) | 204/224 | 2 70 (2 00) | 2.74 (2.05) | 2 47 (2 74) | 2 20 (2 72) | 0.00 |
| mean (sd) | 2.97 (2.65) | 2.75 (2.55) | 3.19 (2.29) | 2.94 (2.24) | 3.78 (2.89) | 3.74 (2.95) | 3.47 (2.71) | 3.38 (2.73) | 0.03 |
| median [IQR] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 3.00 [2.00, 4.00] | 2.00 [1.00, 4.00] | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | 2.79 (2.71) | 2.59 (2.73) | 0.07 |
| Frailty Score (mean): Empirical Version 365 days, | 0.40 (0.07) | 0.47 (0.07) | 0.20 (0.05) | 0.40 (0.00) | 0.24 (0.00) | 0.25 (0.00) | 0.22 (0.07) | 0.22 (0.07) | 2.22 |
| mean (sd) | 0.18 (0.07) | 0.17 (0.07) | 0.20 (0.06) | 0.19 (0.06) | 0.24 (0.08) | 0.25 (0.08) | 0.22 (0.07) | 0.22 (0.07) | 0.00 |
| median [IQR] | 0.17 [0.13, 0.22] | 0.16 [0.12, 0.21] | 0.18 [0.15, 0.22] | 0.18 [0.15, 0.21] | 0.23 [0.19, 0.29] | 0.23 [0.19, 0.29] | 0.21 (0.07) | 0.21 (0.07) | 0.00 |
| Healthcare Utilization | 24 020 (26 | 6 770 /00 000 | 20 526 (20 550) | 44 224 (25 25) | 05 257 (27 650 | 27 777 (26 00() | 454.042.020.200 | 4E 704 (0E 00) | 2.25 |
| Any hospitalization; n (%) | 31,029 (26.4%) | 6,773 (22.8%) | 38,526 (30.9%) | 11,231 (25.9%) | 85,357 (27.9%) | 27,777 (26.8%) | 154,912 (28.2%) | 45,781 (25.9%) | 0.05 |
| Any hospitalization within prior 30 days; n (%) | 14,219 (12.1%) | 2,902 (9.8%) | 16,906 (13.6%) | 4,526 (10.5%) | 33,515 (10.9%) | 10,979 (10.6%) | 64,640 (11.8%) | 18,407 (10.4%) | 0.04 |
| Any hospitalization during prior 31-180 days; n (%) | 19,490 (16.6%) | 4,538 (15.2%) | 24,550 (19.7%) | 7,488 (17.3%) | 60,385 (19.7%) | 19,677 (19.0%) | 104,425 (19.0%) | 31,703 (17.9%) | 0.03 |
| Endocrinologist Visit; n (%) | 7,995 (6.8%) | 3,571 (12.0%) | 8,438 (6.8%) | 5,272 (12.2%) | 25,598 (8.4%) | 13,439 (13.0%) | 42,031 (7.7%) | 22,282 (12.6%) | -0.16 |
| Endocrinologist Visit (30 days prior); n (%) | 4,658 (4.0%) | 2,186 (7.3%) | 5,059 (4.1%) | 3,405 (7.9%) | 13,779 (4.5%) | 7,806 (7.5%) | 23,496 (4.3%) | 13,397 (7.6%) | -0.14 |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 5,356 (4.6%) | 2,429 (8.2%) | 5,416 (4.3%) | 3,438 (7.9%) | 18,906 (6.2%) | 9,468 (9.1%) | 29,678 (5.4%) | 15,335 (8.7%) | -0.13 |
| Internal medicine/family medicine visits; n (%) | 102,084 (86.7%) | 25,865 (86.9%) | 102,764 (82.5%) | 36,903 (85.2%) | 266,343 (87.0%) | 90,264 (87.1%) | 471,191 (85.9%) | 153,032 (86.6%) | -0.02 |
| Internal medicine/family medicine visits (30 days prior); | 76 442 /64 70/ | 10 530 (65 69) | 74 502 (50 000) | 26 002 (62 464) | 100 745 /64 600 | CE CAT (C2 20/) | 220 200 (04 000) | 112.070/02.40() | 0.03 |
| n (%) | 76,112 (64.7%) | 19,520 (65.6%) | 74,503 (59.8%) | 26,903 (62.1%) | 188,745 (61.6%) | 65,647 (63.3%) | 339,360 (61.9%) | 112,070 (63.4%) | -0.03 |

| Internal medicine/family medicine visits (31 to 180 days | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| prior); n (%) | 89,538 (76.1%) | 23,378 (78.6%) | 89,891 (72.1%) | 32,962 (76.1%) | 237,761 (77.6%) | 81,893 (79.0%) | 417,190 (76.0%) | 138,233 (78.2%) | -0.05 |
| Cardiologist visit; n (%) | 64,077 (54.4%) | 16,806 (56.5%) | 57,020 (45.8%) | 21,383 (49.4%) | 183,503 (59.9%) | 63,025 (60.8%) | 304,600 (55.5%) | 101,214 (57.3%) | -0.04 |
| Number of Cardiologist visits (30 days prior); n (%) | 27,683 (23.5%) | 6,944 (23.3%) | 22,417 (18.0%) | 8,351 (19.3%) | 72,663 (23.7%) | 25,568 (24.7%) | 122,763 (22.4%) | 40,863 (23.1%) | -0.02 |
| Number of Conditions in the (21 to 100 down and only of (0/) | F2 002 (44 20/) | 14 115 (47 40/) | 40.005 (20.50/) | 10 177 (42 0%) | 157.007/51.30/\ | E 4 3 E 3 (E 3 30/) | 257 404 (46 0%) | 06 545 (40 0%) | 0.04 |
| Number of Cardiologist visits (31 to 180 days prior); n (%) | 52,002 (44.2%) | 14,115 (47.4%) | 48,005 (38.5%) | 18,177 (42.0%) | 157,097 (51.3%) | 54,253 (52.3%) | 257,104 (46.9%) | 86,545 (49.0%) | -0.04 |
| Electrocardiogram ; n (%) | 60,155 (51.1%) | 15,717 (52.8%) | 62,346 (50.0%) | 22,093 (51.0%) | 168,509 (55.0%) | 59,129 (57.0%) | 291,010 (53.0%) | 96,939 (54.8%) | -0.04 |
| Use of glucose test strips; n (%) | 5,000 (4.2%) | 1,539 (5.2%) | 4,866 (3.9%) | 2,007 (4.6%) | 12,883 (4.2%) | 4,655 (4.5%) | 22,749 (4.1%) | 8,201 (4.6%) | -0.02 |
| Dialysis; n (%) | 775 (0.7%) | 122 (0.4%) | 849 (0.7%) | 225 (0.5%) | 4,837 (1.6%) | 1,196 (1.2%) | 6,461 (1.2%) | 1,543 (0.9%) | 0.03 |
| Naive new user v8 ; n (%) | 49,305 (41.9%) | 10,730 (36.1%) | 51,732 (41.5%) | 15,574 (36.0%) | 110,966 (36.2%) | 33,036 (31.9%) | 212,003 (38.6%) | 59,340 (33.6%) | 0.10 |
| N antidiabetic drugs at index date | | | | | | | | | |
| mean (sd) | 1.52 (0.62) | 1.68 (0.66) | 1.51 (0.63) | 1.67 (0.66) | 1.47 (0.60) | 1.66 (0.66) | 1.49 (0.61) | 1.67 (0.66) | -0.28 |
| median [IQR] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 1.00 (0.61) | 2.00 (0.66) | -1.57 |
| number of different/distinct medication prescriptions | | | | | | | | | |
| mean (sd) | 10.39 (5.16) | 11.20 (5.60) | 10.53 (5.16) | 10.84 (5.32) | 10.98 (5.02) | 11.85 (5.55) | 10.75 (5.08) | 11.49 (5.50) | -0.14 |
| median [IQR] | 10.00 [7.00, 13.00] | 10.00 [7.00, 14.00] | 10.00 [7.00, 13.00] | 10.00 [7.00, 14.00] | 10.00 [7.00, 14.00] | | 10.00 (5.08) | 10.59 (5.50) | -0.14 |
| Number of Hospitalizations | 10.00 [7.00, 13.00] | 10.00 [7.00, 14.00] | 10.00 [7.00, 13.00] | 10.00 [7.00, 14.00] | 10.00 [7.00, 14.00] | .1.00 [8.00, 13.00] | 10.00 (3.08) | 10.55 (5.50) | -0.11 |
| | 0.35 (0.60) | 0.20 (0.05) | 0.20 (0.00) | 0.22 (0.62) | 0.40 (0.77) | 0.20 (0.77) | 0.20 (0.72) | 0.26 (0.72) | 0.04 |
| mean (sd) | 0.35 (0.68) | 0.30 (0.65) | 0.39 (0.68) | 0.32 (0.63) | 0.40 (0.77) | 0.39 (0.77) | 0.39 (0.73) | 0.36 (0.72) | |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.73) | 0.00 (0.72) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 2.18 (6.04) | 1.95 (6.01) | 2.59 (7.05) | 2.15 (6.52) | 2.67 (6.96) | 2.72 (7.33) | 2.55 (6.79) | 2.45 (6.93) | 0.01 |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 3.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 3.00] | 0.00 [0.00, 3.00] | 0.00 (6.79) | 0.00 (6.93) | 0.00 |
| Number of Emergency Department (ED) visits | | | | | | | | | |
| mean (sd) | 0.76 (1.72) | 0.74 (1.78) | 0.59 (2.49) | 0.49 (2.23) | 1.03 (2.00) | 0.98 (2.10) | 0.87 (2.07) | 0.82 (2.08) | 0.02 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 (2.07) | 0.00 (2.08) | 0.00 |
| Number of Office visits | | | | | | | | | |
| mean (sd) | 5.74 (4.68) | 6.30 (4.81) | 6.02 (5.08) | 6.41 (4.84) | 6.56 (5.19) | 7.04 (5.47) | 6.26 (5.06) | 6.76 (5.21) | -0.10 |
| median [IQR] | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 5.00 [3.00, 9.00] | 6.00 [3.00, 10.00] | 5.00 (5.06) | 5.59 (5.21) | -0.11 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.31 (1.81) | 0.59 (2.52) | 0.31 (1.79) | 0.62 (2.88) | 0.46 (2.57) | 0.77 (3.65) | 0.39 (2.26) | 0.70 (3.30) | -0.11 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (2.26) | 0.00 (3.30) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | , | ( , | |
| mean (sd) | 11.67 (16.93) | 11.94 (16.11) | 8.17 (12.67) | 8.75 (12.69) | 10.19 (12.62) | 10.90 (13.48) | 10.05 (13.67) | 10.55 (13.77) | -0.04 |
| median [IQR] | 7.00 [2.00, 15.00] | 7.00 [3.00, 15.00] | 5.00 [1.00, 10.00] | 5.00 [2.00, 11.00] | 6.00 [2.00, 14.00] | , , | 5.99 (13.67) | 6.51 (13.77) | -0.04 |
| Number of Cardiologist visits | 7.00 [2.00, 15.00] | 7.00 [5.00, 15.00] | 5.00 [1.00, 10.00] | 3.00 [2.00, 11.00] | 0.00 [2.00, 14.00] | 7.00 [3.00, 13.00] | 3.33 (13.07) | 0.51 (15.77) | 0.04 |
| mean (sd) | 3.58 (6.52) | 3.72 (6.54) | 2.48 (4.91) | 2.73 (5.15) | 3.71 (6.44) | 3.95 (6.94) | 3.40 (6.14) | 3.61 (6.48) | -0.03 |
| | 1.00 [0.00, 4.00] | 1.00 [0.00, 5.00] | 0.00 [0.00, 3.00] | 0.00 [0.00, 3.00] | | 1.00 [0.00, 5.00] | 0.77 (6.14) | 0.75 (6.48) | 0.00 |
| median [IQR] Number electrocardiograms received | 1.00 [0.00, 4.00] | 1.00 [0.00, 5.00] | 0.00 [0.00, 5.00] | 0.00 [0.00, 5.00] | 1.00 [0.00, 5.00] | 1.00 [0.00, 5.00] | 0.77 (0.14) | 0.73 (0.46) | 0.00 |
| | 1 20 (2 15) | 1 22 (2 27) | 1.00 (1.70) | 1.00 (1.70) | 1 20 (2 02) | 1 42 (2 07) | 1 20 (1 00) | 1 22 (2 02) | -0.02 |
| mean (sd) | 1.28 (2.15) | 1.32 (2.27) | 1.08 (1.70) | 1.08 (1.70) | 1.38 (2.03) | 1.43 (2.07) | 1.29 (1.99) | 1.33 (2.02) | |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 (1.99) | 1.00 (2.02) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 1.04 (0.93) | 1.21 (0.97) | 0.69 (0.87) | 0.83 (0.92) | 1.23 (0.93) | 1.36 (1.00) | 1.07 (0.92) | 1.20 (0.98) | -0.14 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.77 (0.92) | 1.00 (0.98) | -0.24 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.61 (3.51) | 0.82 (5.19) | 0.44 (1.85) | 0.49 (1.71) | 0.49 (1.24) | 0.56 (1.29) | 0.50 (2.07) | 0.59 (2.50) | -0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (2.07) | 0.00 (2.50) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 0.87 (0.99) | 1.04 (1.08) | 0.64 (1.15) | 0.78 (1.21) | 0.92 (0.89) | 1.06 (0.95) | 0.85 (0.98) | 0.99 (1.04) | -0.14 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 0.77 (0.98) | 0.75 (1.04) | 0.02 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.10 (0.50) | 0.10 (0.46) | 0.12 (0.57) | 0.09 (0.44) | 0.15 (0.62) | 0.13 (0.54) | 0.13 (0.58) | 0.12 (0.50) | 0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.58) | 0.00 (0.50) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.07 (0.56) | 0.07 (0.50) | 0.09 (0.57) | 0.07 (0.44) | 0.11 (0.57) | 0.09 (0.49) | 0.10 (0.57) | 0.08 (0.48) | 0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | 0.00 [0.00, 0.00] | 0.00 (0.57) | 0.00 (0.48) | 0.00 |
| Number of tests for microalbuminuria | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 2.23 [0.00, 0.00] | 0.00 (0.57) | 0.00 (0.40) | 0.00 |
| mean (sd) | 0.55 (1.04) | 0.66 (1.15) | 0.31 (0.79) | 0.40 (0.92) | 0.38 (0.72) | 0.43 (0.77) | 0.40 (0.81) | 0.46 (0.88) | -0.07 |
| | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.40 (0.92) | , , | 0.43 (0.77) | 0.00 (0.81) | 0.46 (0.88) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.81) | 0.00 (0.88) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit | | | | | | | | | |
| level | C 02 (0 C2) | 7.24 (10.22) | 2.54/7.20\ | 2 (4 /7 42) | 0.10(11.55) | 0.50/11.00 | 7.25 (40.22) | 7.75 (40.00) | 0.01 |
| mean (sd) | 6.83 (9.63) | 7.34 (10.38) | 3.54 (7.30) | 3.64 (7.42) | 9.10 (11.55) | 9.58 (11.86) | 7.35 (10.32) | 7.75 (10.68) | -0.04 |
| median [IQR] | 4.00 [0.00, 10.00] | 4.00 [0.00, 11.00] | 0.00 [0.00, 4.00] | 0.00 [0.00, 4.00] | 5.00 [0.00, 14.00] | 5.00 [0.00, 15.00] | 3.65 (10.32) | 3.61 (10.68) | 0.00 |
| 11 | 44.005 (44.00) | 2 200 (44 20) | 14.002 (44.20) | 4 522 (40 50) | 20.070.42.77 | 42 454 (42 00) | 67.000 (40.00) | 20 242 (44 500) | 2.22 |
| Use of thiazide; n (%) | 14,035 (11.9%) | 3,360 (11.3%) | 14,093 (11.3%) | 4,532 (10.5%) | 38,970 (12.7%) | 12,451 (12.0%) | 67,098 (12.2%) | 20,343 (11.5%) | 0.02 |
| Use of beta blockers; n (%) | 67,251 (57.1%) | 16,807 (56.5%) | 73,540 (59.0%) | 25,059 (57.9%) | 189,722 (61.9%) | 63,832 (61.6%) | 330,513 (60.2%) | 105,698 (59.8%) | 0.01 |
| Use of calcium channel blockers; n (%) | 36,173 (30.7%) | 9,328 (31.3%) | 37,784 (30.3%) | 12,933 (29.9%) | 108,802 (35.5%) | 37,734 (36.4%) | 182,759 (33.3%) | 59,995 (33.9%) | -0.01 |

Table 1: Sitagliptin vs 2nd Generation Sulfonylureas

#### PS-matched

| | Optum | | MarketScan | | Medic | are | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Reference-2nd | I. | Reference-2nd | | Reference-2nd | | Reference-2nd | POOLED | |
| Variable | Generation SUs | Exposure-Sitagliptin | Generation SUs | Exposure-Sitagliptin | Generation SUs | Exposure-Sitagliptin | Generation SUs | Exposure-Sitagliptin | St. Diff. |
| Number of patients | 29727 | 29727 | 42600 | 42600 | 102411 | 102411 | 174,738 | 174,738 | |
| Age | | | | | | | | | |
| mean (sd) | 69.12 (9.30) | 69.12 (9.34) | 66.33 (10.33) | 66.30 (10.16) | 75.64 (7.48) | 75.65 (7.46) | 72.26 (8.57) | 72.26 (8.52) | 0.00 |
| median [IQR] | 69.00 [62.00, 76.00] | 69.00 [62.00, 76.00] | 64.00 [58.00, 74.00] | 64.00 [59.00, 74.00] | 75.00 [69.00, 81.00] | 75.00 [70.00, 81.00] | 71.30 (8.57) | 71.30 (8.52) | 0.00 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 2,134 (7.2%) | 2,058 (6.9%) | 4,943 (11.6%) | 4,689 (11.0%) | 0 (0.0%) | 0 (0.0%) | 7,077 (4.1%) | 6,747 (3.9%) | 0.01 |
| 55 - 64; n (%) | 7,091 (23.9%) | 7,372 (24.8%) | 17,575 (41.3%) | 17,810 (41.8%) | 1,639 (1.6%) | 1,663 (1.6%) | 26,305 (15.1%) | 26,845 (15.4%) | -0.0 |
| 65 - 74; n (%) | 11,421 (38.4%) | 11,335 (38.1%) | 9,824 (23.1%) | 10,211 (24.0%) | 48,995 (47.8%) | 48,760 (47.6%) | 70,240 (40.2%) | 70,306 (40.2%) | 0.00 |
| >= 75; n (%) | 9,081 (30.5%) | 8,962 (30.1%) | 10,258 (24.1%) | 9,890 (23.2%) | 51,777 (50.6%) | 51,988 (50.8%) | 71,116 (40.7%) | 70,840 (40.5%) | 0.00 |
| Gender- | | | | | | | | | |
| Males; n (%) | 16,707 (56.2%) | 16,770 (56.4%) | 26,043 (61.1%) | 26,160 (61.4%) | 48,955 (47.8%) | 49,246 (48.1%) | 91,705 (52.5%) | 92,176 (52.8%) | -0.01 |
| Females; n (%) | 13,020 (43.8%) | 12,957 (43.6%) | 16,557 (38.9%) | 16,440 (38.6%) | 53,456 (52.2%) | 53,165 (51.9%) | 83,033 (47.5%) | 82,562 (47.2%) | 0.01 |
| Race without zero category | | | | | | | | | |
| White; n (%) | N/A | N/A | N/A | N/A | 78,029 (76.2%) | 78,110 (76.3%) | 78,029 (76.2%) | 78,110 (76.3%) | 0.00 |
| Black; n (%) | N/A | N/A | N/A | N/A | 11,990 (11.7%) | 11,921 (11.6%) | 11,990 (11.7%) | 11,921 (11.6%) | 0.00 |
| Asian; n (%) | N/A | N/A | N/A | N/A | 4,049 (4.0%) | 4,135 (4.0%) | 4,049 (4.0%) | 4,135 (4.0%) | 0.00 |
| Hispanic; n (%) | N/A | N/A | N/A | N/A | 4,455 (4.4%) | 4,419 (4.3%) | 4,455 (4.4%) | 4,419 (4.3%) | 0.00 |
| North American Native; n (%) | N/A | N/A | N/A | N/A | 507 (0.5%) | 527 (0.5%) | 507 (0.5%) | 527 (0.5%) | 0.00 |
| Other/Unknown; n (%) Region- (lumping missing&other category with | N/A | N/A | N/A | N/A | 3,381 (3.3%) | 3,299 (3.2%) | 3,381 (3.3%) | 3,299 (3.2%) | 0.01 |
| West) | | | | | | | | | |
| Northeast; n (%) | 4,282 (14.4%) | 4,214 (14.2%) | 9,061 (21.3%) | 9,017 (21.2%) | 23,934 (23.4%) | 23,883 (23.3%) | 37,277 (21.3%) | 37,114 (21.2%) | 0.00 |
| South; n (%) | 14,991 (50.4%) | 15,045 (50.6%) | 11,460 (26.9%) | 11,433 (26.8%) | 42,802 (41.8%) | 42,665 (41.7%) | 69,253 (39.6%) | 69,143 (39.6%) | 0.00 |
| Midwest; n (%) | 4,983 (16.8%) | 5,055 (17.0%) | 17,261 (40.5%) | 17,306 (40.6%) | 19,090 (18.6%) | 19,020 (18.6%) | 41,334 (23.7%) | 41,381 (23.7%) | 0.00 |
| West; n (%) | 5,471 (18.4%) | 5,413 (18.2%) | 4,420 (10.4%) | 4,425 (10.4%) | 16,585 (16.2%) | 16,843 (16.4%) | 26,476 (15.2%) | 26,681 (15.3%) | 0.00 |
| Unknown+missing; n (%) | N/A | N/A | 398 (0.9%) | 419 (1.0%) | N/A | N/A | 398 (0.9%) | 419 (1.0%) | -0.01 |
| CV Covariates | | | 555 (5.57.) | | | | () | .== (=:=) | |
| Ischemic heart disease; n (%) | 19,747 (66.4%) | 19,742 (66.4%) | 27,261 (64.0%) | 27,300 (64.1%) | 69,177 (67.5%) | 69,239 (67.6%) | 116,185 (66.5%) | 116,281 (66.5%) | 0.00 |
| Acute MI; n (%) | 1,484 (5.0%) | 1,555 (5.2%) | 2,434 (5.7%) | 2,420 (5.7%) | 4,732 (4.6%) | 4,708 (4.6%) | 8,650 (5.0%) | 8,683 (5.0%) | 0.00 |
| ACS/unstable angina; n (%) | 1,542 (5.2%) | 1,607 (5.4%) | 2,448 (5.7%) | 2,483 (5.8%) | 4,573 (4.5%) | 4,651 (4.5%) | 8,563 (4.9%) | 8,741 (5.0%) | 0.00 |
| Old MI; n (%) | 2,812 (9.5%) | 2,811 (9.5%) | 2,027 (4.8%) | 2,046 (4.8%) | 9,882 (9.6%) | 9,759 (9.5%) | 14,721 (8.4%) | 14,616 (8.4%) | 0.00 |
| Stable angina; n (%) | 2,591 (8.7%) | 2,601 (8.7%) | 3,005 (7.1%) | 2,982 (7.0%) | 8,120 (7.9%) | 8,137 (7.9%) | 13,716 (7.8%) | 13,720 (7.9%) | 0.00 |
| Coronary atherosclerosis and other forms of chronic | , ( , | , ( , | .,, | , , | , , , , , | -, - , - , | -, -, -, | -, -, -, | |
| ischemic heart disease; n (%) | 18,771 (63.1%) | 18,846 (63.4%) | 26,077 (61.2%) | 26,181 (61.5%) | 66,512 (64.9%) | 66,608 (65.0%) | 111,360 (63.7%) | 111,635 (63.9%) | 0.00 |
| Other atherosclerosis with ICD10; n (%) | 790 (2.7%) | 858 (2.9%) | 1,074 (2.5%) | 1,092 (2.6%) | 3,628 (3.5%) | 3,676 (3.6%) | 5,492 (3.1%) | 5,626 (3.2%) | -0.03 |
| Previous cardiac procedure (CABG or PTCA or Stent) | | | | | | | | | |
| v4; n (%) | 1,030 (3.5%) | 1,123 (3.8%) | 2,130 (5.0%) | 2,269 (5.3%) | 2,370 (2.3%) | 2,554 (2.5%) | 5,530 (3.2%) | 5,946 (3.4%) | -0.01 |
| History of CABG or PTCA; n (%) | 4,453 (15.0%) | 4,624 (15.6%) | 3,519 (8.3%) | 3,414 (8.0%) | 19,111 (18.7%) | 18,973 (18.5%) | 27,083 (15.5%) | 27,011 (15.5%) | 0.00 |
| Any stroke; n (%) | 6,435 (21.6%) | 6,459 (21.7%) | 8,532 (20.0%) | 8,599 (20.2%) | 25,540 (24.9%) | 25,325 (24.7%) | 40,507 (23.2%) | 40,383 (23.1%) | 0.00 |
| Ischemic stroke (w and w/o mention of cerebral | | | | | | | | | |
| infarction); n (%) | 6,395 (21.5%) | 6,429 (21.6%) | 8,476 (19.9%) | 8,544 (20.1%) | 25,344 (24.7%) | 25,140 (24.5%) | 40,215 (23.0%) | 40,113 (23.0%) | 0.00 |
| Hemorrhagic stroke; n (%) | 153 (0.5%) | 181 (0.6%) | 267 (0.6%) | 269 (0.6%) | 731 (0.7%) | 734 (0.7%) | 1,151 (0.7%) | 1,184 (0.7%) | 0.00 |
| TIA; n (%) | 1,271 (4.3%) | 1,290 (4.3%) | 1,638 (3.8%) | 1,664 (3.9%) | 5,051 (4.9%) | 5,085 (5.0%) | 7,960 (4.6%) | 8,039 (4.6%) | 0.00 |
| Other cerebrovascular disease; n (%) | 1,504 (5.1%) | 1,522 (5.1%) | 1,619 (3.8%) | 1,534 (3.6%) | 6,569 (6.4%) | 6,547 (6.4%) | 9,692 (5.5%) | 9,603 (5.5%) | 0.00 |
| Late effects of cerebrovascular disease; n (%) | 1,537 (5.2%) | 1,504 (5.1%) | 1,428 (3.4%) | 1,404 (3.3%) | 6,846 (6.7%) | 6,639 (6.5%) | 9,811 (5.6%) | 9,547 (5.5%) | 0.00 |
| Cerebrovascular procedure; n (%) | 121 (0.4%) | 95 (0.3%) | 185 (0.4%) | 183 (0.4%) | 347 (0.3%) | 366 (0.4%) | 653 (0.4%) | 644 (0.4%) | 0.00 |
| Heart failure (CHF); n (%) | 5,804 (19.5%) | 5,818 (19.6%) | 6,286 (14.8%) | 6,163 (14.5%) | 24,326 (23.8%) | 24,239 (23.7%) | 36,416 (20.8%) | 36,220 (20.7%) | 0.00 |
| Peripheral Vascular Disease (PVD) or PVD Surgery ; n | | | | | | | | | |
| (%) | 4,609 (15.5%) | 4,584 (15.4%) | 4,885 (11.5%) | 4,787 (11.2%) | 22,088 (21.6%) | 22,005 (21.5%) | 31,582 (18.1%) | 31,376 (18.0%) | 0.00 |
| Atrial fibrillation; n (%) | 4,253 (14.3%) | 4,299 (14.5%) | 5,058 (11.9%) | 5,049 (11.9%) | 21,032 (20.5%) | 20,931 (20.4%) | 30,343 (17.4%) | 30,279 (17.3%) | 0.00 |
| Other cardiac dysrhythmia; n (%) | 5,074 (17.1%) | 5,103 (17.2%) | 5,630 (13.2%) | 5,736 (13.5%) | 23,178 (22.6%) | 23,020 (22.5%) | 33,882 (19.4%) | 33,859 (19.4%) | 0.00 |
| Cardiac conduction disorders; n (%) | 1,629 (5.5%) | 1,675 (5.6%) | 1,733 (4.1%) | 1,742 (4.1%) | 8,051 (7.9%) | 7,876 (7.7%) | 11,413 (6.5%) | 11,293 (6.5%) | 0.00 |
| Other CVD; n (%) | 7,186 (24.2%) | 7,142 (24.0%) | 9,007 (21.1%) | 9,016 (21.2%) | 29,402 (28.7%) | 29,351 (28.7%) | 45,595 (26.1%) | 45,509 (26.0%) | 0.00 |
| Diabetes-related complications | | | | | | | | | |
| Diabetic retinopathy; n (%) | 1,918 (6.5%) | 1,899 (6.4%) | 1,668 (3.9%) | 1,667 (3.9%) | 6,863 (6.7%) | 6,927 (6.8%) | 10,449 (6.0%) | 10,493 (6.0%) | 0.00 |
| Diabetes with other ophthalmic manifestations; n | | | | | | | | | |
| (%) | 167 (0.6%) | 145 (0.5%) | 1,278 (3.0%) | 1,276 (3.0%) | 2,810 (2.7%) | 2,793 (2.7%) | 4,255 (2.4%) | 4,214 (2.4%) | 0.00 |

| Retinal detachment, vitreous hemorrhage, | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| vitrectomy; n (%) | 135 (0.5%) | 149 (0.5%) | 133 (0.3%) | 166 (0.4%) | 425 (0.4%) | 464 (0.5%) | 693 (0.4%) | 779 (0.4%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 182 (0.6%) | 173 (0.6%) | 260 (0.6%) | 284 (0.7%) | 580 (0.6%) | 607 (0.6%) | 1,022 (0.6%) | 1,064 (0.6%) | 0.00 |
| Occurrence of Diabetic Neuropathy; n (%) | 5,913 (19.9%) | 5,840 (19.6%) | 4,816 (11.3%) | 4,778 (11.2%) | 22,008 (21.5%) | 21,921 (21.4%) | 32,737 (18.7%) | 32,539 (18.6%) | 0.00 |
| Occurrence of diabetic nephropathy with ICD10; n | 4 524 (45 20() | 4.40.4 (4.5.40() | 2.452 (5.00() | 2 424 (5 70/) | 44 652 (44 40) | 44 540 (44 20/) | 40.636.(40.70/) | 40 445 (40 50() | 2.24 |
| (%) | 4,521 (15.2%)<br>1,110 (3.7%) | 4,484 (15.1%)<br>1,077 (3.6%) | 2,463 (5.8%)<br>1,283 (3.0%) | 2,421 (5.7%)<br>1,306 (3.1%) | 11,652 (11.4%)<br>4,201 (4.1%) | 11,510 (11.2%)<br>4,170 (4.1%) | 18,636 (10.7%)<br>6,594 (3.8%) | 18,415 (10.5%)<br>6,553 (3.8%) | 0.01<br>0.00 |
| Hypoglycemia; n (%)<br>Hyperglycemia; n (%) | 1,789 (6.0%) | 1,795 (6.0%) | 1,763 (4.1%) | 1,772 (4.2%) | 7,494 (7.3%) | 7,515 (7.3%) | 11,046 (6.3%) | 11,082 (6.3%) | 0.00 |
| Disorders of fluid electrolyte and acid-base balance; n | 1,783 (0.0%) | 1,753 (0.0%) | 1,703 (4.170) | 1,772 (4.270) | 7,434 (7.370) | 7,313 (7.376) | 11,040 (0.376) | 11,082 (0.376) | 0.00 |
| (%) | 3,986 (13.4%) | 4,093 (13.8%) | 3,893 (9.1%) | 3,929 (9.2%) | 17,450 (17.0%) | 17,131 (16.7%) | 25,329 (14.5%) | 25,153 (14.4%) | 0.00 |
| Diabetic ketoacidosis; n (%) | 3 (0.0%) | 4 (0.0%) | 2 (0.0%) | 6 (0.0%) | 31 (0.0%) | 29 (0.0%) | 036 (0.0%) | 039 (0.0%) | #DIV/0! |
| Hyperosmolar hyperglycemic nonketotic syndrome | | | | | | | | | |
| (HONK); n (%) | 180 (0.6%) | 186 (0.6%) | 201 (0.5%) | 207 (0.5%) | 751 (0.7%) | 762 (0.7%) | 1,132 (0.6%) | 1,155 (0.7%) | -0.01 |
| Diabetes with peripheral circulatory disorders with | | | | | | | | | |
| ICD-10 ; n (%) | 2,922 (9.8%) | 2,927 (9.8%) | 2,271 (5.3%) | 2,171 (5.1%) | 11,073 (10.8%) | 11,106 (10.8%) | 16,266 (9.3%) | 16,204 (9.3%) | 0.00 |
| Diabetic Foot; n (%) | 1,120 (3.8%) | 1,127 (3.8%) | 1,347 (3.2%) | 1,292 (3.0%) | 4,785 (4.7%) | 4,658 (4.5%) | 7,252 (4.2%) | 7,077 (4.1%) | 0.01 |
| Gangrene; n (%) | 222 (0.7%)<br>571 (1.9%) | 213 (0.7%)<br>560 (1.9%) | 260 (0.6%)<br>437 (1.0%) | 254 (0.6%)<br>403 (0.9%) | 663 (0.6%)<br>1,712 (1.7%) | 639 (0.6%) | 1,145 (0.7%) | 1,106 (0.6%) | 0.01<br>0.01 |
| Lower extremity amputation; n (%) Osteomyelitis; n (%) | 403 (1.4%) | 399 (1.3%) | 519 (1.2%) | 457 (1.1%) | 1,712 (1.7%) | 1,718 (1.7%)<br>1,267 (1.2%) | 2,720 (1.6%)<br>2,195 (1.3%) | 2,681 (1.5%)<br>2,123 (1.2%) | 0.01 |
| Skin infections ; n (%) | 2,301 (7.7%) | 2,363 (7.9%) | 3,071 (7.2%) | 3,038 (7.1%) | 10,296 (10.1%) | 10,122 (9.9%) | 15,668 (9.0%) | 15,523 (8.9%) | 0.00 |
| Erectile dysfunction; n (%) | 775 (2.6%) | 802 (2.7%) | 888 (2.1%) | 881 (2.1%) | 2,403 (2.3%) | 2,380 (2.3%) | 4,066 (2.3%) | 4,063 (2.3%) | 0.00 |
| Diabetes with unspecified complication; n (%) | 1,863 (6.3%) | 1,849 (6.2%) | 1,859 (4.4%) | 1,814 (4.3%) | 6,426 (6.3%) | 6,351 (6.2%) | 10,148 (5.8%) | 10,014 (5.7%) | 0.00 |
| Diabetes mellitus without mention of complications; | _, | _,_ (=,_,, | _,, | _,, | 5,125 (51571) | 0,000 (0.2) | | | |
| n (%) | 27,552 (92.7%) | 27,521 (92.6%) | 40,513 (95.1%) | 40,470 (95.0%) | 97,729 (95.4%) | 97,734 (95.4%) | 165,794 (94.9%) | 165,725 (94.8%) | 0.00 |
| Hypertension: 1 inpatient or 2 outpatient claims | | | | | | | | | |
| within 365 days; n (%) | 26,771 (90.1%) | 26,773 (90.1%) | 31,437 (73.8%) | 31,407 (73.7%) | 97,195 (94.9%) | 97,173 (94.9%) | 155,403 (88.9%) | 155,353 (88.9%) | 0.00 |
| Hyperlipidemia ; n (%) | 23,855 (80.2%) | 23,797 (80.1%) | 25,697 (60.3%) | 25,671 (60.3%) | 84,137 (82.2%) | 84,130 (82.1%) | 133,689 (76.5%) | 133,598 (76.5%) | 0.00 |
| Edema; n (%) | 3,092 (10.4%) | 3,153 (10.6%) | 2,925 (6.9%) | 2,853 (6.7%) | 15,151 (14.8%) | 15,070 (14.7%) | 21,168 (12.1%) | 21,076 (12.1%) | 0.00 |
| Renal Dysfunction (non-diabetic); n (%) | 8,526 (28.7%) | 8,686 (29.2%) | 7,501 (17.6%) | 7,507 (17.6%) | 33,142 (32.4%) | 32,819 (32.0%) | 49,169 (28.1%) | 49,012 (28.0%) | 0.00 |
| Occurrence of acute renal disease; n (%) | 2,238 (7.5%) | 2,298 (7.7%) | 2,338 (5.5%) | 2,329 (5.5%) | 9,092 (8.9%) | 8,926 (8.7%) | 13,668 (7.8%) | 13,553 (7.8%) | 0.00 |
| Occurrence of chronic renal insufficiency; n (%) | 6,518 (21.9%)<br>6,285 (21.1%) | 6,621 (22.3%)<br>6,406 (21.5%) | 4,835 (11.3%)<br>4,651 (10.9%) | 4,740 (11.1%)<br>4,584 (10.8%) | 25,668 (25.1%)<br>24,388 (23.8%) | 25,291 (24.7%)<br>24,047 (23.5%) | 37,021 (21.2%)<br>35,324 (20.2%) | 36,652 (21.0%)<br>35,037 (20.1%) | 0.00<br>0.00 |
| Chronic kidney disease ; n (%)<br>CKD Stage 3-4; n (%) | 6,285 (21.1%)<br>4,145 (13.9%) | 6,406 (21.5%)<br>4,161 (14.0%) | 4,651 (10.9%)<br>2,852 (6.7%) | 4,584 (10.8%)<br>2,859 (6.7%) | 24,388 (23.8%)<br>15,873 (15.5%) | 24,047 (23.5%)<br>15,739 (15.4%) | 35,324 (20.2%)<br>22,870 (13.1%) | 35,037 (20.1%)<br>22,759 (13.0%) | 0.00 |
| Occurrence of hypertensive nephropathy; n (%) | 3,411 (11.5%) | 3,468 (11.7%) | 2,193 (5.1%) | 2,217 (5.2%) | 13,686 (13.4%) | 13,414 (13.1%) | 19,290 (11.0%) | 19,099 (10.9%) | 0.00 |
| Occurrence of miscellaneous renal insufficiency; n | 3,411 (11.370) | 3,400 (11.770) | 2,133 (3.170) | 2,217 (3.270) | 13,000 (13.470) | 15,414 (15.170) | 13,230 (11.070) | 13,033 (10.370) | 0.00 |
| (%) | 2,817 (9.5%) | 2,845 (9.6%) | 2,640 (6.2%) | 2,693 (6.3%) | 11,951 (11.7%) | 11,930 (11.6%) | 17,408 (10.0%) | 17,468 (10.0%) | 0.00 |
| Glaucoma or cataracts ; n (%) | 5,943 (20.0%) | 6,088 (20.5%) | 7,023 (16.5%) | 7,005 (16.4%) | 26,942 (26.3%) | 27,628 (27.0%) | 39,908 (22.8%) | 40,721 (23.3%) | -0.01 |
| Cellulitis or abscess of toe; n (%) | 631 (2.1%) | 580 (2.0%) | 586 (1.4%) | 604 (1.4%) | 2,291 (2.2%) | 2,264 (2.2%) | 3,508 (2.0%) | 3,448 (2.0%) | 0.00 |
| Foot ulcer; n (%) | 1,138 (3.8%) | 1,125 (3.8%) | 1,380 (3.2%) | 1,322 (3.1%) | 4,839 (4.7%) | 4,694 (4.6%) | 7,357 (4.2%) | 7,141 (4.1%) | 0.01 |
| Bladder stones; n (%) | 50 (0.2%) | 47 (0.2%) | 57 (0.1%) | 57 (0.1%) | 280 (0.3%) | 257 (0.3%) | 387 (0.2%) | 361 (0.2%) | 0.00 |
| Kidney stones; n (%) | 859 (2.9%) | 875 (2.9%) | 1,050 (2.5%) | 1,089 (2.6%) | 3,806 (3.7%) | 3,735 (3.6%) | 5,715 (3.3%) | 5,699 (3.3%) | 0.00 |
| Urinary tract infections (UTIs); n (%) | 3,935 (13.2%) | 3,948 (13.3%) | 3,824 (9.0%) | 3,849 (9.0%) | 22,033 (21.5%) | 21,918 (21.4%) | 29,792 (17.0%) | 29,715 (17.0%) | 0.00 |
| Dipstick urinalysis; n (%) | 11,544 (38.8%) | 12,011 (40.4%) | 13,540 (31.8%) | 13,806 (32.4%) | 48,563 (47.4%) | 49,255 (48.1%) | 73,647 (42.1%) | 75,072 (43.0%) | -0.02 |
| Non-dipstick urinalysis; n (%) | 10,656 (35.8%) | 10,724 (36.1%) | 10,365 (24.3%) | 10,251 (24.1%) | 36,142 (35.3%) | 36,237 (35.4%) | 57,163 (32.7%) | 57,212 (32.7%) | 0.00 |
| Urine function test; n (%) | 1,027 (3.5%)<br>512 (1.7%) | 963 (3.2%)<br>506 (1.7%) | 1,439 (3.4%)<br>942 (2.2%) | 1,533 (3.6%)<br>1,019 (2.4%) | 4,908 (4.8%)<br>2,366 (2.3%) | 5,253 (5.1%)<br>2,440 (2.4%) | 7,374 (4.2%)<br>3,820 (2.2%) | 7,749 (4.4%)<br>3,965 (2.3%) | -0.01<br>-0.01 |
| Cytology; n (%)<br>Cystos; n (%) | 649 (2.2%) | 654 (2.2%) | 1,037 (2.4%) | 1,019 (2.4%) | 3,050 (3.0%) | 2,976 (2.9%) | 4,736 (2.7%) | 4,716 (2.7%) | 0.00 |
| Other Covariates | 043 (2.276) | 034 (2.270) | 1,037 (2.470) | 1,000 (2.570) | 3,030 (3.0%) | 2,370 (2.370) | 4,730 (2.770) | 4,710 (2.776) | 0.00 |
| Liver disease; n (%) | 1,450 (4.9%) | 1,449 (4.9%) | 1,712 (4.0%) | 1,706 (4.0%) | 5,633 (5.5%) | 5,716 (5.6%) | 8,795 (5.0%) | 8,871 (5.1%) | 0.00 |
| Osteoarthritis; n (%) | 5,746 (19.3%) | 5,678 (19.1%) | 5,761 (13.5%) | 5,728 (13.4%) | 29,354 (28.7%) | 29,454 (28.8%) | 40,861 (23.4%) | 40,860 (23.4%) | 0.00 |
| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | |
| pain; n (%) | 13,225 (44.5%) | 13,184 (44.4%) | 15,938 (37.4%) | 15,775 (37.0%) | 57,375 (56.0%) | 57,366 (56.0%) | 86,538 (49.5%) | 86,325 (49.4%) | 0.00 |
| Dorsopathies; n (%) | 7,645 (25.7%) | 7,663 (25.8%) | 8,975 (21.1%) | 9,034 (21.2%) | 33,337 (32.6%) | 33,387 (32.6%) | 49,957 (28.6%) | 50,084 (28.7%) | 0.00 |
| Fractures; n (%) | 1,335 (4.5%) | 1,325 (4.5%) | 1,729 (4.1%) | 1,680 (3.9%) | 6,526 (6.4%) | 6,427 (6.3%) | 9,590 (5.5%) | 9,432 (5.4%) | 0.00 |
| Falls; n (%) | 1,648 (5.5%) | 1,676 (5.6%) | 671 (1.6%) | 669 (1.6%) | 7,999 (7.8%) | 7,998 (7.8%) | 10,318 (5.9%) | 10,343 (5.9%) | 0.00 |
| Osteoporosis; n (%) | 2,026 (6.8%) | 1,959 (6.6%) | 1,826 (4.3%) | 1,829 (4.3%) | 11,401 (11.1%) | 11,491 (11.2%) | 15,253 (8.7%) | 15,279 (8.7%) | 0.00 |
| Hyperthyroidism; n (%) | 258 (0.9%) | 273 (0.9%) | 254 (0.6%) | 269 (0.6%) | 1,392 (1.4%) | 1,291 (1.3%) | 1,904 (1.1%) | 1,833 (1.0%) | 0.01 |
| Hypothyroidism; n (%) | 5,006 (16.8%) | 5,007 (16.8%) | 4,596 (10.8%) | 4,556 (10.7%) | 18,859 (18.4%) | 18,715 (18.3%) | 28,461 (16.3%) | 28,278 (16.2%) | 0.00 |
| Other disorders of thyroid gland; n (%) | 1,304 (4.4%)<br>3,342 (11.2%) | 1,297 (4.4%)<br>3,384 (11.4%) | 1,405 (3.3%)<br>3,165 (7.4%) | 1,511 (3.5%)<br>3,203 (7.5%) | 5,386 (5.3%)<br>16,712 (16.3%) | 5,644 (5.5%)<br>16,568 (16.2%) | 8,095 (4.6%)<br>23,219 (13.3%) | 8,452 (4.8%)<br>23,155 (13.3%) | -0.01<br>0.00 |
| Depression; n (%) Anxiety; n (%) | 3,342 (11.2%)<br>2,701 (9.1%) | 3,384 (11.4%)<br>2,670 (9.0%) | 3,165 (7.4%)<br>2,053 (4.8%) | 3,203 (7.5%)<br>2,071 (4.9%) | 16,712 (16.3%) | 16,568 (16.2%) | 23,219 (13.3%)<br>17,466 (10.0%) | 23,155 (13.3%)<br>17,307 (9.9%) | 0.00 |
| Sleep_Disorder; n (%) | 3,198 (10.8%) | 3,169 (10.7%) | 4,986 (11.7%) | 4,912 (11.5%) | 12,712 (12.4%) | 12,566 (12.3%) | 17,466 (10.0%) | 17,307 (9.9%) | 0.00 |
| Dementia; n (%) | 2,224 (7.5%) | 2,267 (7.6%) | 1,970 (4.6%) | 1,919 (4.5%) | 14,941 (14.6%) | 14,723 (14.4%) | 19,135 (11.0%) | 18,909 (10.8%) | 0.01 |
| Delirium; n (%) | 884 (3.0%) | 914 (3.1%) | 984 (2.3%) | 996 (2.3%) | 5,202 (5.1%) | 5,036 (4.9%) | 7,070 (4.0%) | 6,946 (4.0%) | 0.00 |
| Psychosis; n (%) | 582 (2.0%) | 615 (2.1%) | 598 (1.4%) | 593 (1.4%) | 4,032 (3.9%) | 3,917 (3.8%) | 5,212 (3.0%) | 5,125 (2.9%) | 0.01 |
| Obesity; n (%) | 5,273 (17.7%) | 5,251 (17.7%) | 4,452 (10.5%) | 4,430 (10.4%) | 16,002 (15.6%) | 15,920 (15.5%) | 25,727 (14.7%) | 25,601 (14.7%) | 0.00 |
| Overweight; n (%) | 1,301 (4.4%) | 1,275 (4.3%) | 597 (1.4%) | 604 (1.4%) | 3,724 (3.6%) | 3,738 (3.6%) | 5,622 (3.2%) | 5,617 (3.2%) | 0.00 |

| C | 4,679 (15.7%) | 4,679 (15.7%) | 3,092 (7.3%) | 3,132 (7.4%) | 19,687 (19.2%) | 19,521 (19.1%) | 27,458 (15.7%) | 27,332 (15.6%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Smoking; n (%) | 4,679 (15.7%)<br>287 (1.0%) | 4,679 (15.7%)<br>287 (1.0%) | 3,092 (7.3%)<br>264 (0.6%) | 266 (0.6%) | 19,687 (19.2%) | 19,521 (19.1%)<br>899 (0.9%) | 1,438 (0.8%) | 1,452 (0.8%) | 0.00 |
| Alcohol abuse or dependence; n (%) Drug abuse or dependence; n (%) | 453 (1.5%) | 473 (1.6%) | 281 (0.7%) | 259 (0.6%) | 1,406 (1.4%) | 1,440 (1.4%) | 2,140 (1.2%) | 2,172 (1.2%) | 0.00 |
| COPD; n (%) | 4,606 (15.5%) | 4,680 (15.7%) | 4,833 (11.3%) | 4,849 (11.4%) | 19,771 (19.3%) | 19,860 (19.4%) | 29,210 (16.7%) | 29,389 (16.8%) | 0.00 |
| Asthma; n (%) | 2,066 (6.9%) | 2,129 (7.2%) | 2,217 (5.2%) | 2,218 (5.2%) | 8,593 (8.4%) | 8,606 (8.4%) | 12,876 (7.4%) | 12,953 (7.4%) | 0.00 |
| | | | | | | | | | 0.00 |
| Obstructive sleep apnea; n (%) | 3,164 (10.6%) | 3,100 (10.4%) | 4,205 (9.9%) | 4,193 (9.8%) | 9,119 (8.9%) | 9,049 (8.8%) | 16,488 (9.4%) | 16,342 (9.4%) | 0.00 |
| Pneumonia; n (%) | 1,627 (5.5%) | 1,654 (5.6%) | 2,255 (5.3%) | 2,217 (5.2%) | 7,732 (7.5%) | 7,674 (7.5%) | 11,614 (6.6%) | 11,545 (6.6%) | |
| Imaging; n (%) | 146 (0.5%) | 128 (0.4%) | 101 (0.2%) | 114 (0.3%) | 500 (0.5%) | 545 (0.5%) | 747 (0.4%) | 787 (0.5%) | -0.01 |
| Diabetes Medications | 05 (0.20() | 06 (0.20() | 426 (0.20() | 422 (0.20() | 444 (0.40() | 44.4 (0.40() | C 4 2 (0 40() | C 4 2 (D 40() | 0.00 |
| DM Medications - AGIs; n (%) | 96 (0.3%) | 96 (0.3%) | 136 (0.3%) | 133 (0.3%) | 411 (0.4%) | 414 (0.4%) | 643 (0.4%) | 643 (0.4%) | 0.00 |
| DM Medications - Glitazones; n (%) | 2,692 (9.1%) | 2,696 (9.1%) | 4,523 (10.6%) | 4,386 (10.3%) | 5,892 (5.8%) | 5,851 (5.7%) | 13,107 (7.5%) | 12,933 (7.4%) | 0.00 |
| DM Medications - GLP-1 RA; n (%) | 198 (0.7%) | 190 (0.6%) | 182 (0.4%) | 187 (0.4%) | 354 (0.3%) | 332 (0.3%) | #VALUE! | #VALUE! | #VALUE! |
| DM Medications - Insulin; n (%) | 5,880 (19.8%) | 5,819 (19.6%) | 6,527 (15.3%) | 6,474 (15.2%) | 22,926 (22.4%) | 22,323 (21.8%) | 35,333 (20.2%) | 34,616 (19.8%) | 0.01 |
| DM Medications - Meglitinides; n (%) | 577 (1.9%) | 659 (2.2%) | 1,311 (3.1%) | 1,333 (3.1%) | 2,582 (2.5%) | 2,736 (2.7%) | 4,470 (2.6%) | 4,728 (2.7%) | -0.01 |
| DM Medications - Metformin; n (%) | 17,034 (57.3%) | 17,021 (57.3%) | 24,802 (58.2%) | 24,873 (58.4%) | 56,177 (54.9%) | 56,075 (54.8%) | 98,013 (56.1%) | 97,969 (56.1%) | 0.00 |
| Concomitant initiation or current use of SGLT2i; n | | | | | | | | | |
| (%) | 429 (1.4%) | 433 (1.5%) | 501 (1.2%) | 524 (1.2%) | 1,159 (1.1%) | 1,179 (1.2%) | 2,089 (1.2%) | 2,136 (1.2%) | 0.00 |
| Concomitant initiation or current use of AGIs; n (%) | 61 (0.2%) | 64 (0.2%) | 95 (0.2%) | 89 (0.2%) | 289 (0.3%) | 289 (0.3%) | 445 (0.3%) | 442 (0.3%) | 0.00 |
| Concomitant initiation or current use of Glitazones; | 1 457 (4 00/) | 1 440 (4 00/) | 2 200 (5 00/) | 2 200 (5 20/) | 2 257 (2 20/) | 2 200 (2 20/) | 7 102 (4 10/) | 7.000 (4.00/) | 0.01 |
| n (%) Concomitant initiation or current use of GLP-1 RA; n | 1,457 (4.9%) | 1,440 (4.8%) | 2,368 (5.6%) | 2,260 (5.3%) | 3,357 (3.3%) | 3,309 (3.2%) | 7,182 (4.1%) | 7,009 (4.0%) | 0.01 |
| (%) | 70 (0.2%) | 67 (0.2%) | 55 (0.1%) | 57 (0.1%) | 119 (0.1%) | 111 (0.1%) | 244 (0.1%) | 235 (0.1%) | 0.00 |
| | 70 (0.2%) | 67 (0.2%) | 33 (0.1%) | 37 (0.1%) | 119 (0.1%) | 111 (0.176) | 244 (0.1%) | 255 (0.1%) | 0.00 |
| Concomitant initiation or current use of Insulin; n (%) | 3,960 (13.3%) | 3,969 (13.4%) | 4,274 (10.0%) | 4,170 (9.8%) | 15,825 (15.5%) | 15,444 (15.1%) | 24,059 (13.8%) | 23,583 (13.5%) | 0.01 |
| Concomitant initiation or current use of | 3,900 (13.3%) | 3,909 (13.4%) | 4,274 (10.0%) | 4,170 (9.6%) | 13,023 (13.3%) | 13,444 (13.176) | 24,039 (13.6%) | 23,363 (13.3%) | 0.01 |
| Meglitinides; n (%) | 316 (1.1%) | 475 (1.6%) | 746 (1.8%) | 939 (2.2%) | 1,784 (1.7%) | 1,940 (1.9%) | 2,846 (1.6%) | 3,354 (1.9%) | -0.02 |
| Concomitant initiation or current use of Metformin; | 310 (1.1%) | 473 (1.070) | 740 (1.870) | 333 (2.270) | 1,704 (1.770) | 1,340 (1.370) | 2,840 (1.070) | 3,334 (1.370) | -0.02 |
| n (%) | 13,532 (45.5%) | 13,632 (45.9%) | 20,013 (47.0%) | 20,149 (47.3%) | 43,913 (42.9%) | 43,951 (42.9%) | 77,458 (44.3%) | 77,732 (44.5%) | 0.00 |
| Past use of SGLT2i; n (%) | 215 (0.7%) | 209 (0.7%) | 212 (0.5%) | 20,149 (47.5%) | 582 (0.6%) | 43,931 (42.9%)<br>557 (0.5%) | 1,009 (0.6%) | 969 (0.6%) | 0.00 |
| * * * | , , | , , | , , | , , | , , | | | , , | |
| Past use of AGIs; n (%) | 35 (0.1%) | 32 (0.1%) | 41 (0.1%) | 44 (0.1%) | 122 (0.1%) | 125 (0.1%) | 198 (0.1%) | 201 (0.1%) | 0.00 |
| Past use of Glitazones ; n (%) | 1,235 (4.2%) | 1,256 (4.2%) | 2,156 (5.1%) | 2,126 (5.0%) | 2,535 (2.5%) | 2,542 (2.5%) | 5,926 (3.4%) | 5,924 (3.4%) | 0.00 |
| Past use of GLP-1 RA; n (%) | 131 (0.4%) | 124 (0.4%) | 129 (0.3%) | 133 (0.3%) | 235 (0.2%) | 221 (0.2%) | 495 (0.3%) | 478 (0.3%) | 0.00 |
| Past use of Insulin ; n (%) | 1,920 (6.5%) | 1,850 (6.2%) | 2,253 (5.3%) | 2,305 (5.4%) | 7,103 (6.9%) | 6,882 (6.7%) | 11,276 (6.5%) | 11,037 (6.3%) | 0.01 |
| Past use of Meglitinides ; n (%) | 261 (0.9%) | 184 (0.6%) | 565 (1.3%) | 394 (0.9%) | 798 (0.8%) | 796 (0.8%) | 1,624 (0.9%) | 1,374 (0.8%) | 0.01 |
| Past use of metformin (final); n (%) | 3,502 (11.8%) | 3,389 (11.4%) | 4,789 (11.2%) | 4,724 (11.1%) | 12,264 (12.0%) | 12,124 (11.8%) | 20,555 (11.8%) | 20,237 (11.6%) | 0.01 |
| Other Medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 12,130 (40.8%) | 12,196 (41.0%) | 17,833 (41.9%) | 17,824 (41.8%) | 40,301 (39.4%) | 40,254 (39.3%) | 70,264 (40.2%) | 70,274 (40.2%) | 0.00 |
| Use of ARBs; n (%) | 8,377 (28.2%) | 8,297 (27.9%) | 12,003 (28.2%) | 12,003 (28.2%) | 31,904 (31.2%) | 31,978 (31.2%) | 52,284 (29.9%) | 52,278 (29.9%) | 0.00 |
| Use of Loop Diuretics - ; n (%) | 6,654 (22.4%) | 6,700 (22.5%) | 8,970 (21.1%) | 8,915 (20.9%) | 29,451 (28.8%) | 29,240 (28.6%) | 45,075 (25.8%) | 44,855 (25.7%) | 0.00 |
| Use of other diuretics-; n (%) | 1,482 (5.0%) | 1,460 (4.9%) | 2,026 (4.8%) | 2,032 (4.8%) | 5,716 (5.6%) | 5,595 (5.5%) | 9,224 (5.3%) | 9,087 (5.2%) | 0.00 |
| Use of nitrates-; n (%) | 4,156 (14.0%) | 4,225 (14.2%) | 6,759 (15.9%) | 6,740 (15.8%) | 16,769 (16.4%) | 16,892 (16.5%) | 27,684 (15.8%) | 27,857 (15.9%) | 0.00 |
| Use of other hypertension drugs; n (%) | 2,725 (9.2%) | 2,775 (9.3%) | 3,435 (8.1%) | 3,452 (8.1%) | 11,247 (11.0%) | 11,238 (11.0%) | 17,407 (10.0%) | 17,465 (10.0%) | 0.00 |
| Use of digoxin-; n (%) | 1,243 (4.2%) | 1,265 (4.3%) | 2,096 (4.9%) | 2,094 (4.9%) | 5,653 (5.5%) | 5,682 (5.5%) | 8,992 (5.1%) | 9,041 (5.2%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | 1,009 (3.4%) | 1,037 (3.5%) | 1,646 (3.9%) | 1,637 (3.8%) | 4,512 (4.4%) | 4,398 (4.3%) | 7,167 (4.1%) | 7,072 (4.0%) | 0.01 |
| Use of COPD/asthma meds-; n (%) | 5,314 (17.9%) | 5,331 (17.9%) | 7,511 (17.6%) | 7,445 (17.5%) | 22,193 (21.7%) | 22,356 (21.8%) | 35,018 (20.0%) | 35,132 (20.1%) | 0.00 |
| Use of statins; n (%) | 21,217 (71.4%) | 21,259 (71.5%) | 30,505 (71.6%) | 30,420 (71.4%) | 74,884 (73.1%) | 74,789 (73.0%) | 126,606 (72.5%) | 126,468 (72.4%) | 0.00 |
| Use of other lipid-lowering drugs; n (%) | 4,653 (15.7%) | 4,636 (15.6%) | 8,222 (19.3%) | 8,219 (19.3%) | 14,426 (14.1%) | 14,315 (14.0%) | 27,301 (15.6%) | 27,170 (15.5%) | 0.00 |
| Use of antiplatelet agents; n (%) | 8,723 (29.3%) | 8,787 (29.6%) | 14,464 (34.0%) | 14,420 (33.8%) | 29,939 (29.2%) | 30,180 (29.5%) | 53,126 (30.4%) | 53,387 (30.6%) | 0.00 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, | | | | | | | | | |
| Apixaban, Warfarin); n (%) | 3,349 (11.3%) | 3,375 (11.4%) | 4,638 (10.9%) | 4,669 (11.0%) | 15,605 (15.2%) | 15,554 (15.2%) | 23,592 (13.5%) | 23,598 (13.5%) | 0.00 |
| Use of heparin and other low-molecular weight | | | | | | | | | |
| heparins; n (%) | 266 (0.9%) | 249 (0.8%) | 36 (0.1%) | 31 (0.1%) | 932 (0.9%) | 931 (0.9%) | 1,234 (0.7%) | 1,211 (0.7%) | 0.00 |
| Use of NSAIDs; n (%) | 4,026 (13.5%) | 4,031 (13.6%) | 5,599 (13.1%) | 5,656 (13.3%) | 16,708 (16.3%) | 16,790 (16.4%) | 26,333 (15.1%) | 26,477 (15.2%) | 0.00 |
| Use of oral corticosteroids; n (%) | 5,138 (17.3%) | 5,237 (17.6%) | 7,511 (17.6%) | 7,423 (17.4%) | 22,295 (21.8%) | 22,282 (21.8%) | 34,944 (20.0%) | 34,942 (20.0%) | 0.00 |
| Use of bisphosphonate (); n (%) | 939 (3.2%) | 924 (3.1%) | 1,106 (2.6%) | 1,119 (2.6%) | 4,332 (4.2%) | 4,362 (4.3%) | 6,377 (3.6%) | 6,405 (3.7%) | -0.01 |
| Use of opioids-; n (%) | 9,061 (30.5%) | 9,112 (30.7%) | 13,177 (30.9%) | 13,185 (31.0%) | 32,771 (32.0%) | 32,800 (32.0%) | 55,009 (31.5%) | 55,097 (31.5%) | 0.00 |
| Use of antidepressants; n (%) | 7,899 (26.6%) | 7,878 (26.5%) | 10,404 (24.4%) | 10,233 (24.0%) | 31,518 (30.8%) | 31,530 (30.8%) | 49,821 (28.5%) | 49,641 (28.4%) | 0.00 |
| Use of antipsychotics; n (%) | 982 (3.3%) | 988 (3.3%) | 1,038 (2.4%) | 994 (2.3%) | 5,625 (5.5%) | 5,472 (5.3%) | 7,645 (4.4%) | 7,454 (4.3%) | 0.00 |
| Use of anticonvulsants; n (%) | 5,309 (17.9%) | 5,312 (17.9%) | 6,020 (14.1%) | 5,899 (13.8%) | 22,554 (22.0%) | 22,494 (22.0%) | 33,883 (19.4%) | 33,705 (19.3%) | 0.00 |
| Use of lithium- ; n (%) | 49 (0.2%) | 46 (0.2%) | 64 (0.2%) | 62 (0.1%) | 169 (0.2%) | 124 (0.1%) | 282 (0.2%) | 232 (0.1%) | 0.03 |
| Use of Benzos- ; n (%) | 3,328 (11.2%) | 3,370 (11.3%) | 5,785 (13.6%) | 5,788 (13.6%) | 13,195 (12.9%) | 13,059 (12.8%) | 22,308 (12.8%) | 22,217 (12.7%) | 0.00 |
| Use of anxiolytics/hypnotics-; n (%) | 2,212 (7.4%) | 2,250 (7.6%) | 3,697 (8.7%) | 3,609 (8.5%) | 8,941 (8.7%) | 9,025 (8.8%) | 14,850 (8.5%) | 14,884 (8.5%) | 0.00 |
| Use of dementia meds-; n (%) | 1,145 (3.9%) | 1,142 (3.8%) | 1,201 (2.8%) | 1,199 (2.8%) | 8,554 (8.4%) | 8,470 (8.3%) | 10,900 (6.2%) | 10,811 (6.2%) | 0.00 |
| | | | | | | | | | 0.00 |
| Use of antiparkinsonian meds-; n (%) | 875 (2.9%) | 915 (3.1%) | 1,237 (2.9%) | 1,176 (2.8%) | 4,679 (4.6%) | 4,656 (4.5%) | 6,791 (3.9%) | 6,747 (3.9%) | |
| Any use of pramlintide; n (%) | 8 (0.0%) | 9 (0.0%) | 28 (0.1%) | 37 (0.1%) | 12 (0.0%) | 27 (0.0%) | 048 (0.0%) | 073 (0.0%) | #DIV/0! |
| Any use of 1st generation sulfonylureas; n (%) | 15 (0.1%) | 11 (0.0%) | 41 (0.1%) | 15 (0.0%) | 51 (0.0%) | 27 (0.0%) | 107 (0.1%) | 053 (0.0%) | 0.00 |
| Entresto (sacubitril/valsartan); n (%) | 56 (0.2%) | 65 (0.2%) | 23 (0.1%) | 19 (0.0%) | 93 (0.1%) | 120 (0.1%) | 172 (0.1%) | 204 (0.1%) | 0.00 |

| Initiation as monotherapy v4 ; n (%) | 7,093 (23.9%) | 7,240 (24.4%) | 9,995 (23.5%) | 10,304 (24.2%) | 20,129 (19.7%) | 20,714 (20.2%) | 37,217 (21.3%) | 38,258 (21.9%) | -0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Labs | | | | | | | 72,327 | 72,327 | |
| Lab values- HbA1c (%); n (%) | 8,669 (29.2%) | 8,827 (29.7%) | 2,042 (4.8%) | 1,847 (4.3%) | N/A | N/A | 10,711 (14.8%) | 10,674 (14.8%) | 0.00 |
| Lab values- HbA1c (%) (within 3 months); n (%) | 6,595 (22.2%) | 6,705 (22.6%) | 1,575 (3.7%) | 1,424 (3.3%) | N/A | N/A | 8,170 (11.3%) | 8,129 (11.2%) | 0.00 |
| Lab values- HbA1c (%) (within 6 months); n (%) | 8,669 (29.2%) | 8,827 (29.7%) | 2,042 (4.8%) | 1,847 (4.3%) | N/A | N/A | 10,711 (14.8%) | 10,674 (14.8%) | 0.00 |
| Lab values- BNP; n (%) | 329 (1.1%) | 354 (1.2%) | 66 (0.2%) | 73 (0.2%) | N/A | N/A | 395 (0.5%) | 427 (0.6%) | -0.01 |
| Lab values- BNP (within 3 months); n (%) | 201 (0.7%) | 219 (0.7%) | 42 (0.1%) | 54 (0.1%) | N/A | N/A | 243 (0.3%) | 273 (0.4%) | -0.02 |
| Lab values- BNP (within 6 months); n (%) | 329 (1.1%) | 354 (1.2%) | 66 (0.2%) | 73 (0.2%) | N/A | N/A | 395 (0.5%) | 427 (0.6%) | -0.01 |
| Lab values- BUN (mg/dl); n (%) | 9,465 (31.8%) | 9,769 (32.9%) | 1,999 (4.7%) | 2,034 (4.8%) | N/A | N/A | 11,464 (15.9%) | 11,803 (16.3%) | -0.01 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 7,205 (24.2%) | 7,482 (25.2%) | 1,527 (3.6%) | 1,550 (3.6%) | N/A | N/A | 8,732 (12.1%) | 9,032 (12.5%) | -0.01 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 9,465 (31.8%) | 9,769 (32.9%) | 1,999 (4.7%) | 2,034 (4.8%) | N/A | N/A | 11,464 (15.9%) | 11,803 (16.3%) | -0.01 |
| Lab values- Creatinine (mg/dl); n (%) | 9,694 (32.6%) | 10,013 (33.7%) | 2,137 (5.0%) | 2,158 (5.1%) | N/A | N/A | 11,831 (16.4%) | 12,171 (16.8%) | -0.01 |
| Lab values- Creatinine (mg/dl) (within 3 months); n | | | | | | | | | |
| (%) | 7,384 (24.8%) | 7,681 (25.8%) | 1,642 (3.9%) | 1,636 (3.8%) | N/A | N/A | 9,026 (12.5%) | 9,317 (12.9%) | -0.01 |
| Lab values- Creatinine (mg/dl) (within 6 months); n | | | | | | | | | |
| (%) | 9,694 (32.6%) | 10,013 (33.7%) | 2,137 (5.0%) | 2,158 (5.1%) | N/A | N/A | 11,831 (16.4%) | 12,171 (16.8%) | -0.01 |
| Lab values- HDL level (mg/dl); n (%) | 7,615 (25.6%) | 7,857 (26.4%) | 1,837 (4.3%) | 1,684 (4.0%) | N/A | N/A | 9,452 (13.1%) | 9,541 (13.2%) | 0.00 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 5,408 (18.2%) | 5,644 (19.0%) | 1,322 (3.1%) | 1,239 (2.9%) | N/A | N/A | 6,730 (9.3%) | 6,883 (9.5%) | -0.01 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 7,615 (25.6%) | 7,857 (26.4%) | 1,837 (4.3%) | 1,684 (4.0%) | N/A | N/A | 9,452 (13.1%) | 9,541 (13.2%) | 0.00 |
| Lab values- LDL level (mg/dl) ; n (%) | 7,779 (26.2%) | 8,047 (27.1%) | 1,951 (4.6%) | 1,792 (4.2%) | N/A | N/A<br>N/A | 9,730 (13.5%) | 9,839 (13.6%) | 0.00 |
| Lab values- LDL level (Hig/GI) , II (76) | 7,773 (20.270) | 8,047 (27.178) | 1,331 (4.0%) | 1,732 (4.270) | N/A | IN/A | 3,730 (13.370) | 3,833 (13.0%) | 0.00 |
| Lab values- LDL level (mg/dl) (within 3 months); n (%) | 5,526 (18.6%) | 5,768 (19.4%) | 1,406 (3.3%) | 1,317 (3.1%) | N/A | N/A | 6,932 (9.6%) | 7,085 (9.8%) | -0.01 |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 7,779 (26.2%) | 8,047 (27.1%) | 1,951 (4.6%) | 1,792 (4.2%) | N/A | N/A | 9,730 (13.5%) | 9,839 (13.6%) | 0.00 |
| Lab values- NT-proBNP; n (%) | 46 (0.2%) | 43 (0.1%) | 3 (0.0%) | 3 (0.0%) | N/A | N/A | 49 (0.1%) | 0 (0.1%) | - |
| Lab values- NT-proBNP (within 3 months); n (%) | 28 (0.1%) | 19 (0.1%) | 2 (0.0%) | 2 (0.0%) | N/A | N/A | 30 (0.0%) | 0 (0.0%) | - |
| Lab values- NT-proBNP (within 6 months); n (%) | 46 (0.2%) | 43 (0.1%) | 3 (0.0%) | 3 (0.0%) | N/A | N/A | 49 (0.1%) | 46 (0.1%) | - |
| Lab values-Total cholesterol (mg/dl); n (%) | 7,723 (26.0%) | 7,976 (26.8%) | 1,908 (4.5%) | 1,761 (4.1%) | N/A | N/A | 9,631 (13.3%) | 9,737 (13.5%) | -0.01 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | |
| months); n (%) | 5,490 (18.5%) | 5,723 (19.3%) | 1,373 (3.2%) | 1,289 (3.0%) | N/A | N/A | 6,863 (9.5%) | 7,012 (9.7%) | -0.01 |
| Lab values- Total cholesterol (mg/dl) (within 6 | 7 722 (25 00() | 7.076 (26.00() | 4 000 (4 50() | 4.764 (4.40) | | 21/2 | 0.624 (42.20() | 0.727 (42.50) | -0.01 |
| months); n (%) | 7,723 (26.0%) | 7,976 (26.8%) | 1,908 (4.5%) | 1,761 (4.1%) | N/A | N/A | 9,631 (13.3%) | 9,737 (13.5%) | |
| Lab values-Triglyceride level (mg/dl); n (%) | 7,638 (25.7%) | 7,867 (26.5%) | 1,873 (4.4%) | 1,730 (4.1%) | N/A | N/A | 9,511 (13.1%) | 9,597 (13.3%) | -0.01 |
| Lab values-Triglyceride level (mg/dl) (within 3 months); n (%) | 5,426 (18.3%) | 5,641 (19.0%) | 1,351 (3.2%) | 1,273 (3.0%) | N/A | N/A | 6,777 (9.4%) | 6,914 (9.6%) | -0.01 |
| Lab values-Triglyceride level (mg/dl) (within 6 | 3,420 (18.5%) | 3,041 (19.0%) | 1,331 (3.2%) | 1,273 (5.0%) | IN/A | IN/A | 6,777 (9.4%) | 0,914 (9.0%) | -0.01 |
| months); n (%) | 7,638 (25.7%) | 7,867 (26.5%) | 1,873 (4.4%) | 1,730 (4.1%) | N/A | N/A | 9,511 (13.1%) | 9,597 (13.3%) | -0.01 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | 7,030 (23.770) | 7,007 (20.570) | 1,073 (4.470) | 1,730 (4.170) | 14/15 | 14/7 | 5,511 (15.170) | 3,337 (13.370) | 0.01 |
| included) v4 | 8,595 | 8,741 | 1,872 | 1,782 | N/A | N/A | 10,467 | 10,523 | |
| mean (sd) | 7.99 (1.78) | 7.78 (1.69) | 8.13 (1.88) | 7.90 (1.75) | N/A | N/A | 8.02 (1.80) | 7.80 (1.70) | 0.13 |
| median [IQR] | 7.60 [6.80, 8.80] | 7.40 [6.60, 8.50] | 7.70 [6.80, 9.00] | 7.45 [6.70, 8.65] | N/A | N/A | 7.62 (1.80) | 7.41 (1.70) | 0.12 |
| Missing; n (%) | 21,132 (71.1%) | 20,986 (70.6%) | 40,728 (95.6%) | 40,818 (95.8%) | N/A | N/A | 61,860 (85.5%) | 61,804 (85.5%) | 0.00 |
| Lab result number- BNP mean | 329 | 354 | 66 | 73 | N/A | N/A | 395 | 427 | |
| mean (sd) | 221.45 (330.00) | 212.58 (353.05) | 324.29 (602.41) | 213.53 (315.86) | N/A | N/A | 238.63 (388.97) | 212.74 (347.44) | 0.07 |
| median [IQR] | 97.00 [38.70, 238.45] | 106.60 [36.45, 239.20] | 89.50 [29.62, 339.62] | 101.00 [32.00, 264.25] | N/A | N/A | #VALUE! | 105.64 (347.44) | #VALUE! |
| Missing; n (%) | 29,398 (98.9%) | 29,373 (98.8%) | 42,534 (99.8%) | 42,527 (99.8%) | N/A | N/A | 71,932 (99.5%) | 71,900 (99.4%) | 0.01 |
| Lab result number- BUN (mg/dl) mean | 9,465 | 9,769 | 1,999 | 2,034 | N/A | N/A | 11,464 | 11,803 | |
| mean (sd) | 20.54 (9.90) | 20.26 (9.38) | 844.91 (11,853.76) | 221.96 (5,038.61) | N/A | N/A | 164.29 (4949.29) | 55.02 (2091.42) | 0.03 |
| median [IQR] | 18.00 [14.00, 24.00] | 18.00 [14.00, 23.77] | 17.00 [14.00, 22.00] | 17.00 [14.00, 22.00] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 20,262 (68.2%) | 19,958 (67.1%) | 40,601 (95.3%) | 40,566 (95.2%) | N/A | N/A | 60,863 (84.1%) | 60,524 (83.7%) | 0.01 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | | | | | | | | | |
| to 15 included) | 9,619 | 9,904 | 2,042 | 2,033 | N/A | N/A | 11,661 | 11,937 | |
| mean (sd) | 1.13 (0.55) | 1.13 (0.55) | 1.07 (0.59) | 1.05 (0.51) | N/A | N/A | 1.12 (0.56) | 1.12 (0.54) | 0.00 |
| median [IQR] | 1.01 [0.83, 1.29] | 1.02 [0.84, 1.28] | 0.98 [0.80, 1.16] | 0.98 [0.81, 1.15] | N/A | N/A | 1.00 (0.56) | 1.01 (0.54) | -0.02 |
| Missing; n (%) | 20,108 (67.6%) | 19,823 (66.7%) | 40,558 (95.2%) | 40,567 (95.2%) | N/A | N/A | 60,666 (83.9%) | 60,390 (83.5%) | 0.01 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | |
| =<5000 included) | 7,615 | 7,857 | 1,830 | 1,683 | N/A | N/A | 9,445 | 9,540 | |
| mean (sd) | 44.85 (13.87) | 45.38 (14.01) | 43.92 (15.63) | 43.57 (14.19) | N/A | N/A | 44.67 (14.23) | 45.06 (14.04) | -0.03 |
| median [IQR] | 43.00 [36.00, 52.00] | 44.00 [36.00, 53.00] | 42.00 [35.00, 51.00] | 42.00 [35.00, 51.00] | N/A | N/A | 42.81 (14.23) | 43.65 (14.04) | -0.06 |
| Missing; n (%) | 22,112 (74.4%) | 21,870 (73.6%) | 40,770 (95.7%) | 40,917 (96.0%) | N/A | N/A | 62,882 (86.9%) | 62,787 (86.8%) | 0.00 |
| Lab result number- LDL level (mg/dl) mean (only | 7.617 | 7.005 | 4.004 | 1.694 | N/A | N/A | 9.441 | 9.579 | |
| =<5000 included) | 7,617<br>85.26 (40.77) | 7,885<br>83.19 (39.97) | 1,824 | *** | N/A<br>N/A | | | | 0.05 |
| mean (sd)<br>median [IQR] | 85.26 (40.77)<br>82.00 [61.00, 109.00] | 83.19 (39.97)<br>79.40 [59.00, 104.00] | 87.55 (41.77)<br>85.00 [62.50, 112.00] | 86.51 (42.89)<br>83.00 [62.00, 111.00] | N/A<br>N/A | N/A<br>N/A | 85.70 (40.97)<br>82.58 (40.97) | 83.78 (40.50)<br>80.04 (40.50) | 0.05 |
| | 22,110 (74.4%) | 21,842 (73.5%) | 40,776 (95.7%) | 40,906 (96.0%) | N/A<br>N/A | N/A<br>N/A | 62,886 (86.9%) | 80.04 (40.50)<br>62,748 (86.8%) | 0.06 |
| Missing; n (%) | 22,110 (74.4%) | 21,042 (/3.5%) | 40,770 (33.7%) | 40,500 (50.0%) | IN/A | IN/A | 02,000 (00.3%) | 02,740 (00.0%) | 0.00 |

| Lab result number-Total cholesterol (mg/dl) mean | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (only =<5000 included) | 7,718 | 7,965 | 1,900 | 1,757 | N/A | N/A | 9,618 | 9,722 | |
| mean (sd) | 170.55 (48.85) | 167.26 (48.37) | 172.88 (50.42) | 171.42 (51.31) | N/A | N/A | 171.01 (49.17) | 168.01 (48.92) | 0.06 |
| median [IQR] | 164.00 [138.00, 197.00] | 161.00 [136.50, 191.50] | 167.00 [142.00, 199.00] | 166.00 [140.00, 198.00] | N/A | N/A | 164.59 (49.17) | 161.90 (48.92) | 0.05 |
| Missing; n (%) | 22,009 (74.0%) | 21,762 (73.2%) | 40,700 (95.5%) | 40,843 (95.9%) | N/A | N/A | 62,709 (86.7%) | 62,605 (86.6%) | 0.00 |
| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | | | |
| (only =<5000 included) | 7,638 | 7,867 | 1,866 | 1,729 | N/A | N/A | 9,504 | 9,596 | |
| mean (sd) | 187.28 (156.16) | 178.93 (148.77) | 189.86 (160.62) | 191.36 (174.88) | N/A | N/A | 187.79 (157.05) | 181.17 (153.81) | 0.04 |
| median [IQR] | 152.00 [109.00, 215.00] | | 152.00 [106.38, 218.50] | 149.33 [106.25, 219.00] | N/A | N/A | 152.00 (157.05) | 146.60 (153.81) | 0.03 |
| Missing; n (%) | 22,089 (74.3%) | 21,860 (73.5%) | 40,734 (95.6%) | 40,871 (95.9%) | N/A | N/A | 62,823 (86.9%) | 62,731 (86.7%) | 0.01 |
| Lab result number- Hemoglobin mean (only >0 | | | | | | | | | |
| included) | 7,029 | 7,205 | 1,467 | 1,399 | N/A | N/A | 8,496 | 8,604 | |
| mean (sd) | 13.26 (1.79) | 13.26 (1.76) | 612.63 (9,372.79) | 321.61 (6,152.32) | N/A | N/A | 116.75 (3894.08) | 63.40 (2480.38) | 0.02 |
| median [IQR] | 13.30 [12.10, 14.50] | 13.30 [12.10, 14.50] | 13.50 [12.30, 14.70] | 13.50 [12.30, 14.70] | N/A | N/A | #VALUE! | #VALUE! | #VALUE! |
| Missing; n (%) | 22,698 (76.4%) | 22,522 (75.8%) | 41,133 (96.6%) | 41,201 (96.7%) | N/A | N/A | 63,831 (88.3%) | 63,723 (88.1%) | 0.01 |
| Lab result number- Serum sodium mean (only > 90 | | | | | | | | | |
| and < 190 included) | 9,400 | 9,693 | 1,874 | 1,847 | N/A | N/A | 11,274 | 11,540 | |
| mean (sd) | 139.35 (2.89) | 139.52 (2.83) | 138.98 (2.87) | 139.11 (2.74) | N/A | N/A | 139.29 (2.89) | 139.45 (2.82) | -0.06 |
| median [IQR] | 139.50 [138.00, 141.00] | | 139.00 [137.50, 141.00] | 139.00 [137.50, 141.00] | N/A | N/A | 139.42 (2.89) | 139.84 (2.82) | -0.15 |
| Missing; n (%) | 20,327 (68.4%) | 20,034 (67.4%) | 40,726 (95.6%) | 40,753 (95.7%) | N/A | N/A | 61,053 (84.4%) | 60,787 (84.0%) | 0.01 |
| Lab result number- Albumin mean (only >0 and <=10 included) | 8,711 | 9,009 | 1,706 | 1,663 | N/A | N/A | 10,417 | 10,672 | |
| • | 4.17 (0.35) | 4.17 (0.35) | 4.15 (0.52) | 4.14 (0.59) | N/A<br>N/A | N/A | 4.17 (0.38) | 4.17 (0.40) | 0.00 |
| mean (sd)<br>median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.43] | N/A<br>N/A | N/A | 4.20 (0.38) | 4.20 (0.40) | 0.00 |
| Missing; n (%) | 21,016 (70.7%) | 20,718 (69.7%) | 40,894 (96.0%) | 40,937 (96.1%) | N/A<br>N/A | N/A | 61,910 (85.6%) | 61,655 (85.2%) | 0.00 |
| Lab result number- Glucose (fasting or random) mean | 21,010 (70.7%) | 20,710 (09.7%) | 40,694 (90.0%) | 40,937 (90.1%) | N/A | IN/A | 01,910 (03.0%) | 01,033 (83.2%) | 0.01 |
| (only 10-1000 included) | 9,394 | 9,695 | 1,867 | 1,826 | N/A | N/A | 11,261 | 11,521 | |
| mean (sd) | 168.15 (72.56) | 161.26 (67.24) | 173.78 (76.66) | 164.94 (72.28) | N/A | N/A | 169.08 (73.26) | 161.84 (68.07) | 0.10 |
| median [IQR] | 150.00 [121.00, 195.50] | 144.00 [117.00, 185.00] | 153.67 [124.00, 202.50] | 145.00 [119.00, 189.00] | N/A | N/A | 150.61 (73.26) | 144.16 (68.07) | 0.09 |
| Missing; n (%) | 20,333 (68.4%) | 20,032 (67.4%) | 40,733 (95.6%) | 40,774 (95.7%) | N/A | N/A | 61,066 (84.4%) | 60,806 (84.1%) | 0.01 |
| Lab result number- Potassium mean (only 1-7 | 20,555 (60:170) | 20,032 (07.170) | 10,755 (55.070) | 10,771 (33.770) | .,,,, | | 01,000 (0 11 170) | 00,000 (0 1.170) | 0.01 |
| included) | 9,573 | 9,878 | 1,980 | 1,995 | N/A | N/A | 11,553 | 11,873 | |
| mean (sd) | 4.45 (0.45) | 4.43 (0.45) | 4.37 (0.44) | 4.38 (0.44) | N/A | N/A | 4.44 (0.45) | 4.42 (0.45) | 0.04 |
| median [IQR] | 4.40 [4.15, 4.70] | 4.40 [4.12, 4.70] | 4.35 [4.05, 4.70] | 4.40 [4.10, 4.65] | N/A | N/A | 4.39 (0.45) | 4.40 (0.45) | -0.02 |
| Missing; n (%) | 20,154 (67.8%) | 19,849 (66.8%) | 40,620 (95.4%) | 40,605 (95.3%) | N/A | N/A | 60,774 (84.0%) | 60,454 (83.6%) | 0.01 |
| Comorbidity Scores | ., . ( , | .,, | ., ( , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , | , | , , | , . (, | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 3.53 (2.31) | 3.54 (2.35) | 2.57 (2.10) | 2.56 (2.12) | 4.21 (2.40) | 4.19 (2.41) | 3.69 (2.31) | 3.68 (2.33) | 0.00 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 4.00 [2.00, 6.00] | 4.00 [2.00, 6.00] | 3.34 (2.31) | 3.34 (2.33) | 0.00 |
| Frailty Score: Qualitative Version 365 days as | | | | | | | | | |
| Categories, v1 | | | | | | | | | |
| 0; n (%) | 6,384 (21.5%) | 5,865 (19.7%) | 3,424 (8.0%) | 3,464 (8.1%) | 15,773 (15.4%) | 15,429 (15.1%) | 25,581 (14.6%) | 24,758 (14.2%) | 0.01 |
| 1 to 2; n (%) | 10,115 (34.0%) | 10,511 (35.4%) | 18,141 (42.6%) | 18,211 (42.7%) | 24,197 (23.6%) | 24,350 (23.8%) | 52,453 (30.0%) | 53,072 (30.4%) | -0.01 |
| 3 or more; n (%) | 13,228 (44.5%) | 13,351 (44.9%) | 21,035 (49.4%) | 20,925 (49.1%) | 62,441 (61.0%) | 62,632 (61.2%) | 96,704 (55.3%) | 96,908 (55.5%) | 0.00 |
| Frailty Score: Empirical Version 365 days as | | | | | | | | | |
| Categories, | | | | | | | | | |
| <0.12908; n (%) | 1,610 (5.4%) | 1,675 (5.6%) | 2,733 (6.4%) | 2,919 (6.9%) | 1,887 (1.8%) | 2,260 (2.2%) | 6,230 (3.6%) | 6,854 (3.9%) | -0.02 |
| 0.12908 - 0.1631167; n (%) | 6,451 (21.7%) | 6,526 (22.0%) | 10,144 (23.8%) | 10,347 (24.3%) | 10,000 (9.8%) | 10,659 (10.4%) | 26,595 (15.2%) | 27,532 (15.8%) | -0.02 |
| >= 0.1631167; n (%) | 21,666 (72.9%) | 21,526 (72.4%) | 29,723 (69.8%) | 29,334 (68.9%) | 90,524 (88.4%) | 89,492 (87.4%) | 141,913 (81.2%) | 140,352 (80.3%) | 0.02 |
| Non-Frailty; n (%) | 16,772 (56.4%) | 16,976 (57.1%) | 21,481 (50.4%) | 21,489 (50.4%) | 3,954 (3.9%) | 3,683 (3.6%) | 42,207 (24.2%) | 42,148 (24.1%) | 0.00 |
| Fully Country to the | | | | | | | | | |
| Frailty Score (mean): Qualitative Version 365 days, v1 | 2 74 (2 55) | 2.75 (2.55) | 2.05 (2.22) | 2.05 (2.24) | 2 72 (2 04) | 2.72 (2.05) | 2 26 (2 72) | 2 27 (2 72) | 2.00 |
| mean (sd) | 2.71 (2.55)<br>2.00 [1.00, 4.00] | 2.75 (2.55)<br>2.00 [1.00, 4.00] | 2.95 (2.22) | 2.95 (2.24)<br>2.00 [1.00, 4.00] | 3.72 (2.94)<br>3.00 [1.00, 6.00] | 3.73 (2.95)<br>3.00 [1.00, 6.00] | 3.36 (2.72) | 3.37 (2.73)<br>2.59 (2.73) | 0.00<br>0.00 |
| median [IQR] Frailty Score (mean): Empirical Version 365 days, | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | 2.59 (2.72) | 2.59 (2.73) | 0.00 |
| | 0.17 (0.07) | 0.17 (0.07) | 0.19 (0.06) | 0.19 (0.06) | 0.25 (0.08) | 0.25 (0.08) | 0.22 (0.07) | 0.22 (0.07) | 0.00 |
| mean (sd)<br>median [IQR] | 0.16 [0.12, 0.21] | 0.16 [0.12, 0.21] | 0.18 [0.15, 0.22] | 0.18 [0.15, 0.21] | 0.23 [0.19, 0.29] | 0.23 [0.19, 0.29] | 0.21 (0.07) | 0.22 (0.07) | 0.00 |
| Healthcare Utilization | 0.10 [0.12, 0.21] | 0.10 [0.12, 0.21] | 0.18 [0.13, 0.22] | 0.18 [0.13, 0.21] | 0.23 [0.13, 0.23] | 0.23 [0.13, 0.23] | 0.21 (0.07) | 0.21 (0.07) | 0.00 |
| Any hospitalization; n (%) | 6,882 (23.2%) | 6,765 (22.8%) | 11,065 (26.0%) | 11,100 (26.1%) | 27,916 (27.3%) | 27,495 (26.8%) | 45,863 (26.2%) | 45,360 (26.0%) | 0.00 |
| Any hospitalization, it (%) Any hospitalization within prior 30 days; n (%) | 2,859 (9.6%) | 2,900 (9.8%) | 4,437 (10.4%) | 4,490 (10.5%) | 10,985 (10.7%) | 10,851 (10.6%) | 18,281 (10.5%) | 18,241 (10.4%) | 0.00 |
| Any hospitalization within prior 30 days, ir (%) Any hospitalization during prior 31-180 days; n (%) | 4,537 (15.3%) | 4,531 (15.2%) | 7,362 (17.3%) | 7,387 (17.3%) | 19,769 (19.3%) | 19,486 (19.0%) | 31,668 (18.1%) | 31,404 (18.0%) | 0.00 |
| Endocrinologist Visit; n (%) | 3,404 (11.5%) | 3,551 (11.9%) | 4,825 (11.3%) | 4,946 (11.6%) | 12,520 (12.2%) | 12,940 (12.6%) | 20,749 (11.9%) | 21,437 (12.3%) | -0.01 |
| Endocrinologist Visit, i1 (%) Endocrinologist Visit (30 days prior); n (%) | 2,140 (7.2%) | 2,169 (7.3%) | 3,180 (7.5%) | 3,140 (7.4%) | 7,592 (7.4%) | 7,411 (7.2%) | 12,912 (7.4%) | 12,720 (7.3%) | 0.00 |
| Endocrinologist Visit (30 days prior), it (%) Endocrinologist Visit (31 to 180 days prior); it (%) | 2,399 (8.1%) | 2,412 (8.1%) | 3,183 (7.5%) | 3,140 (7.4%) | 9,156 (8.9%) | 9,098 (8.9%) | 14,738 (8.4%) | 14,705 (8.4%) | 0.00 |
| Internal medicine/family medicine visits; n (%) | 26,096 (87.8%) | 25,836 (86.9%) | 36,484 (85.6%) | 36,277 (85.2%) | 89,704 (87.6%) | 89,135 (87.0%) | 152,284 (87.1%) | 151,248 (86.6%) | 0.00 |
| Internal medicine/family medicine visits (30 days | 20,000 (07.070) | 25,050 (00.576) | 30,707 (03.0%) | 30,211 (03.270) | 33,. 34 (07.070) | 03,233 (07.070) | 102,207 (07.170) | 131,2 70 (00.070) | 0.01 |
| prior); n (%) | 19,588 (65.9%) | 19,501 (65.6%) | 26,797 (62.9%) | 26,480 (62.2%) | 64,921 (63.4%) | 64,807 (63.3%) | 111,306 (63.7%) | 110,788 (63.4%) | 0.01 |

| Internal medicine/family medicine visits (31 to 180 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| days prior) ; n (%) | 23,320 (78.4%) | 23,349 (78.5%) | 32,491 (76.3%) | 32,370 (76.0%) | 81,075 (79.2%) | 80,830 (78.9%) | 136,886 (78.3%) | 136,549 (78.1%) | 0.00 |
| Cardiologist visit; n (%) | 16,806 (56.5%) | 16,784 (56.5%) | 21,071 (49.5%) | 20,964 (49.2%) | 62,396 (60.9%) | 62,201 (60.7%) | 100,273 (57.4%) | 99,949 (57.2%) | 0.00 |
| Number of Cardiologist visits (30 days prior); n (%) | 6,841 (23.0%) | 6,934 (23.3%) | 8,260 (19.4%) | 8,178 (19.2%) | 25,354 (24.8%) | 25,197 (24.6%) | 40,455 (23.2%) | 40,309 (23.1%) | 0.00 |
| Number of Cardiologist visits (31 to 180 days prior);<br>n (%) | 14,105 (47.4%) | 14,093 (47.4%) | 17,962 (42.2%) | 17,810 (41.8%) | 53,633 (52.4%) | 53,527 (52.3%) | 85,700 (49.0%) | 85,430 (48.9%) | 0.00 |
| Electrocardiogram ; n (%) | 15,569 (52.4%) | 15,698 (52.8%) | 21,582 (50.7%) | 21,691 (50.9%) | 58,001 (56.6%) | 58,332 (57.0%) | 95,152 (54.5%) | 95,721 (54.8%) | -0.01 |
| Use of glucose test strips; n (%) | 1,526 (5.1%) | 1,536 (5.2%) | 1,947 (4.6%) | 1,947 (4.6%) | 4,540 (4.4%) | 4,587 (4.5%) | 8,013 (4.6%) | 8,070 (4.6%) | 0.00 |
| Dialysis; n (%) | 143 (0.5%) | 122 (0.4%) | 209 (0.5%) | 225 (0.5%) | 1,302 (1.3%) | 1,191 (1.2%) | 1,654 (0.9%) | 1,538 (0.9%) | 0.00 |
| Naive new user v8 ; n (%) | 10,615 (35.7%) | 10,728 (36.1%) | 15,150 (35.6%) | 15,436 (36.2%) | 32,363 (31.6%) | 32,876 (32.1%) | 58,128 (33.3%) | 59,040 (33.8%) | -0.01 |
| N antidiabetic drugs at index date | | | | | | | | | |
| mean (sd) | 1.67 (0.68) | 1.68 (0.66) | 1.66 (0.67) | 1.66 (0.65) | 1.65 (0.67) | 1.65 (0.65) | 1.66 (0.67) | 1.66 (0.65) | 0.00 |
| median [IQR] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | 2.00 (0.67) | 2.00 (0.65) | 0.00 |
| number of different/distinct medication | | | | | | | | | |
| prescriptions | 44 47 (5 40) | 44.40 (5.50) | 40.07 (5.26) | 40.02 (5.24) | 44.04 (5.25) | 44.70 (5.40) | 44.47 (5.25) | 44.45 (5.46) | 2.00 |
| mean (sd) | 11.17 (5.48)<br>10.00 [7.00, 14.00] | 11.19 (5.59)<br>10.00 [7.00, 14.00] | 10.87 (5.26)<br>10.00 [7.00, 14.00] | 10.82 (5.31) | 11.81 (5.35)<br>11.00 [8.00, 15.00] | 11.79 (5.49)<br>11.00 [8.00, 15.00] | 11.47 (5.35) | 11.45 (5.46)<br>10.59 (5.46) | 0.00<br>0.00 |
| median [IQR] Number of Hospitalizations | 10.00 [7.00, 14.00] | 10.00 [7.00, 14.00] | 10.00 [7.00, 14.00] | 10.00 [7.00, 14.00] | 11.00 [8.00, 15.00] | 11.00 [8.00, 15.00] | 10.59 (5.35) | 10.59 (5.46) | 0.00 |
| mean (sd) | 0.30 (0.62) | 0.30 (0.65) | 0.32 (0.62) | 0.32 (0.63) | 0.40 (0.77) | 0.39 (0.77) | 0.36 (0.71) | 0.36 (0.72) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.71) | 0.00 (0.72) | 0.00 |
| Number of hospital days | | | | | | | , | , | |
| mean (sd) | 1.90 (5.67) | 1.95 (6.01) | 2.18 (6.63) | 2.16 (6.53) | 2.78 (7.68) | 2.72 (7.30) | 2.48 (7.12) | 2.45 (6.91) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 3.00] | 0.00 [0.00, 3.00] | 0.00 (7.12) | 0.00 (6.91) | 0.00 |
| Number of Emergency Department (ED) visits | | | | | | | | | |
| mean (sd) | 0.73 (1.64) | 0.74 (1.78) | 0.49 (2.08) | 0.49 (2.24) | 0.99 (1.84) | 0.98 (2.11) | 0.82 (1.87) | 0.82 (2.09) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 (1.87) | 0.00 (2.09) | 0.00 |
| Number of Office visits | 6 20 (4 05) | C 20 (4 00) | C 42 (5 54) | 6 20 (4 00) | C 00 (5 50) | C 00 (5 42) | 6.72 (5.44) | 6 72 (5 47) | 0.00 |
| mean (sd) | 6.28 (4.95) | 6.29 (4.80) | 6.42 (5.51) | 6.38 (4.80) | 6.99 (5.50) | 6.99 (5.42) | 6.73 (5.41) | 6.72 (5.17) | 0.00<br>0.00 |
| median [IQR] Number of Endocrinologist visits | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 6.00 [3.00, 10.00] | 6.00 [3.00, 10.00] | 5.59 (5.41) | 5.59 (5.17) | 0.00 |
| mean (sd) | 0.56 (2.48) | 0.58 (2.51) | 0.54 (2.42) | 0.58 (2.79) | 0.71 (3.34) | 0.74 (3.52) | 0.64 (3.00) | 0.67 (3.20) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (3.00) | 0.00 (3.20) | 0.00 |
| Number of internal medicine/family medicine visits | (,) | (,) | (,) | (,) | (,, | ,, | () | 5.55 (5.25) | |
| mean (sd) | 12.02 (17.25) | 11.94 (16.11) | 8.50 (12.80) | 8.74 (12.71) | 10.70 (13.45) | 10.86 (13.42) | 10.39 (14.02) | 10.53 (13.75) | -0.01 |
| median [IQR] | 7.00 [3.00, 15.00] | 7.00 [3.00, 15.00] | 5.00 [2.00, 11.00] | 5.00 [2.00, 11.00] | 7.00 [3.00, 14.00] | 7.00 [3.00, 15.00] | 6.51 (14.02) | 6.51 (13.75) | 0.00 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 3.60 (6.45) | 3.71 (6.54) | 2.70 (5.12) | 2.72 (5.14) | 3.91 (6.81) | 3.95 (6.94) | 3.56 (6.38) | 3.61 (6.48) | -0.01 |
| median [IQR] | 1.00 [0.00, 5.00] | 1.00 [0.00, 5.00] | 0.00 [0.00, 3.00] | 0.00 [0.00, 3.00] | 1.00 [0.00, 5.00] | 1.00 [0.00, 5.00] | 0.76 (6.38) | 0.76 (6.48) | 0.00 |
| Number electrocardiograms received | 4 20 (2 47) | 4 22 (2 27) | 4.00 (4.67) | 4 00 (4 74) | 4.44(2.00) | 4 42 (2 07) | 4 22 (2 04) | 4 22 (2 02) | 0.00 |
| mean (sd)<br>median [IQR] | 1.29 (2.17)<br>1.00 [0.00, 2.00] | 1.32 (2.27)<br>1.00 [0.00, 2.00] | 1.08 (1.67) | 1.08 (1.71)<br>1.00 [0.00, 1.00] | 1.44 (2.09)<br>1.00 [0.00, 2.00] | 1.43 (2.07) | 1.33 (2.01)<br>1.00 (2.01) | 1.33 (2.03) | 0.00 |
| Number of HbA1c tests ordered | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 1.00 (2.01) | 1.00 (2.03) | 0.00 |
| mean (sd) | 1.21 (0.99) | 1.21 (0.96) | 0.83 (0.94) | 0.82 (0.92) | 1.36 (1.00) | 1.35 (0.99) | 1.21 (0.98) | 1.20 (0.97) | 0.01 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 1.00 (0.98) | 1.00 (0.97) | 0.00 |
| Number of glucose tests ordered | | | | | | | , , | , , | |
| mean (sd) | 0.79 (5.17) | 0.82 (5.19) | 0.50 (1.97) | 0.49 (1.71) | 0.55 (1.41) | 0.55 (1.28) | 0.58 (2.58) | 0.58 (2.50) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (2.58) | 0.00 (2.50) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 1.04 (1.10) | 1.04 (1.07) | 0.79 (1.32) | 0.78 (1.20) | 1.05 (0.96) | 1.05 (0.94) | 0.98 (1.08) | 0.98 (1.03) | 0.00 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.76 (1.08) | 0.76 (1.03) | 0.00 |
| Number of creatinine tests ordered | 0.40 (0.53) | 0.40 (0.46) | 0.10 (0.40) | 0.00 (0.44) | 0.14(0.50) | 0.13 (0.54) | 0.13 (0.55) | 0.13 (0.50) | 0.00 |
| mean (sd)<br>median [IQR] | 0.10 (0.53)<br>0.00 [0.00, 0.00] | 0.10 (0.46)<br>0.00 [0.00, 0.00] | 0.10 (0.48)<br>0.00 [0.00, 0.00] | 0.09 (0.44)<br>0.00 [0.00, 0.00] | 0.14 (0.59)<br>0.00 [0.00, 0.00] | 0.13 (0.54)<br>0.00 [0.00, 0.00] | 0.12 (0.55)<br>0.00 (0.55) | 0.12 (0.50)<br>0.00 (0.50) | 0.00<br>0.00 |
| Number of BUN tests ordered | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.33) | 0.00 (0.50) | 0.00 |
| mean (sd) | 0.07 (0.57) | 0.07 (0.50) | 0.07 (0.48) | 0.07 (0.44) | 0.10 (0.53) | 0.09 (0.49) | 0.09 (0.53) | 0.08 (0.48) | 0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 (0.53) | 0.00 (0.48) | 0.00 |
| Number of tests for microalbuminuria | | | | | | | | | |
| mean (sd) | 0.67 (1.16) | 0.66 (1.15) | 0.40 (0.90) | 0.40 (0.91) | 0.43 (0.78) | 0.43 (0.76) | 0.46 (0.88) | 0.46 (0.87) | 0.00 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.88) | 0.00 (0.87) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | |
| digit level | | | | | | | | | |
| mean (sd) | 7.34 (10.04)<br>4.00 [0.00, 11.00] | 7.34 (10.38)<br>4.00 [0.00, 11.00] | 3.62 (7.39) | 3.63 (7.40) | 9.68 (11.90) | 9.57 (11.86) | 7.80 (10.65)<br>4.20 (10.65) | 7.74 (10.68) | 0.01<br>0.06 |
| median [IQR] | 4.00 [0.00, 11.00] | 4.00 [0.00, 11.00] | 0.00 [0.00, 4.00] | 0.00 [0.00, 4.00] | 6.00 [0.00, 15.00] | 5.00 [0.00, 15.00] | 4.20 (10.05) | 3.61 (10.68) | 0.06 |
| Use of thiazide; n (%) | 3,428 (11.5%) | 3,358 (11.3%) | 4,478 (10.5%) | 4,470 (10.5%) | 12,338 (12.0%) | 12,334 (12.0%) | 20,244 (11.6%) | 20,162 (11.5%) | 0.00 |
| Use of beta blockers; n (%) | 16,752 (56.4%) | 16,787 (56.5%) | 24,718 (58.0%) | 24,658 (57.9%) | 63,213 (61.7%) | 63,051 (61.6%) | 104,683 (59.9%) | 104,496 (59.8%) | 0.00 |
| Use of calcium channel blockers; n (%) | 9,269 (31.2%) | 9,316 (31.3%) | 12,735 (29.9%) | 12,730 (29.9%) | 37,118 (36.2%) | 37,223 (36.3%) | 59,122 (33.8%) | 59,269 (33.9%) | 0.00 |